

# STATISTICAL ANALYSIS PLAN

| Protocol Title | A Multicenter, Randomized, Active-controlled Study to Evaluate the Efficacy and Safety of EXPAREL When Administered via Infiltration into the Transversus Abdominis Plane (TAP) Versus Standard of Care in Subjects Undergoing Elective Cesarean Section. |
|---|---|
| Protocol Number | 402-C-414 |
| Protocol Version | Final |
| Protocol Date | Original: 16 August 2018 Amendment 1: 15Nov2018. Amendment 2: 07 February 2019 |
| Study Drug | EXPAREL (bupivacaine liposome injectable suspension) |
| Study Phase | 4 |
| IND Number | 069,198 |
| Sponsor | Pacira Pharmaceuticals, Inc. 5 Sylvan Way Parsippany, NJ 07054 Tel: 973-254-3560 |
| SAP Version | 1.0 |
| Date | 16 March 2020 |

Pacira Pharmaceuticals, Inc.  $\mathsf{EXPAREL}^{\$}$ 

402-C-414 (C-section TAP) Statistical Analysis Plan

# 1 SIGNATURE PAGE

| Alfred Mbali | 18-Mar-2020 |
|-------------------------------------------------|-------------|
| Alfred Mbah, PhD | Date |
| Principal Statitician | |
| Pharma Data Asociates, LLC | |
| Chao Wang | 17-Mar-2020 |
| Chao Wang, PhD | Date |
| Principal Statitician | |
| Pharma Data Asociates, LLC | |
| Vinant Yu | 17-Mar-2020 |
| Vincent Yu, PhD | Date |
| Vice President, Biometrics | |
| Pacira Pharmaceuticals, Inc | |
| Alla Nagaer | 17-Mar-2020 |
| Alla Nagaev, MD | Date |
| Associate Medical Director, Clinical Operations | |
| Pacira Pharmaceuticals, Inc | |
| Julia Yang | 18-Mar-2020 |
| Julia Yang, MD | Date |
| VP, Clinical Research Pacira | |
| Pharmaceuticals, Inc | |
| Michael Kozycki | 17-Mar-2020 |
| Michael Rozycki, PhD | <br>Date |
| Senior Vice President, Regulatory Affairs | |
| Pacira Pharmaceuticals, Inc | |

402-C-414 (C-section TAP) Statistical Analysis Plan

# 2 TABLE OF CONTENTS

| l | SIGNATURE PAGE | 2 |
|---|---|---|
| 2 | TABLE OF CONTENTS | 3 |
| 3 | LIST OF ABBREVIATIONS | 5 |
| 1 | INTRODUCTION | 6 |
| 5 | STUDY OBJECTIVES | 7 |
| 5.1 | Primary Objective | 7 |
| 5.2 | Secondary Objectives | 7 |
| 6 | STUDY OVERVIEW | 7 |
| 7 | DEFINITIONS | 8 |
| 3 | ANALYSIS SETS | 10 |
| 3.1 | Safety set | 10 |
| 3.2 | Efficacy set | 10 |
| 3.3 | Sensitivity set | 10 |
| ) | STUDY ENDPOINTS | 10 |
| 9.1 | Efficacy Endpoints | 10 |
| 9.1.1 | Primary Efficacy | 10 |
| 9.1.2 | Key Secondary Efficacy | 10 |
| 9.1.3 | Secondary Efficacy | 10 |
| 9.1.4 | Exploratory Efficacy | 11 |
| 9.2 | Safety Endpoints | 11 |
| 9.3 | Efficacy Assessment | 11 |
| 9.3.1 | Opioid Dose Conversion | 11 |
| 9.3.2 | Average Postsurgical VAS pain Intensity Scores Through 72 Hours or Hospital Discharge, Whichever Occurs First. | 12 |
| 9.3.3 | Opioid Related Symptom Distress Scale (ORSDS) | 13 |
| 9.3.4 | Subject Satisfaction with Pain | 13 |
| 9.3.5 | Pain Surgical Fear Questionnaire (SFQ) | 14 |
| 9.3.6 | Pain Calls to Physician (Single Question) | 14 |
| 9.3.7 | Persistent Opioid Use | 14 |
| 9.3.8 | Recovery from Caesarean Section Scale (RCSS) | 14 |
| 10 | STATISTICAL METHODS OF ANALYSIS | 14 |
| 10.1 | General Principles | 14 |
| 0.1.1 | Handling Missing Values | 15 |
| 0.1.1.1 | Total Postsurgery Opioid Consumption | 15 |


| Pacira Phar<br>EXPAREL® | 402-C-414 (C-section TAP)<br>Statistical Analysis Plan | |
|---|---|---|
| 10.1.1.2 | Postsurgical Itching Scores through 72 hours | 15 |
| 10.1.1.3 | VAS Pain Intensity Scores | 15 |
| 10.1.1.4 | Exposure, Surgery, and Rescue Medication Date or Time | 16 |
| 10.1.1.5 | Adverse Event or Concomitant Medications Dates or Times | 16 |
| 10.1.1.6 | Adverse Event Severity or Relationship to Study Drug | 16 |
| 10.1.1.7 | Time to Event | 17 |
| 10.1.2 | By-Center Analyses | 17 |
| 10.1.3 | Non-Inferiority Margin (NIM) | 17 |
| 10.2 | Subject Disposition | 17 |
| 10.3 | Description of Demographics and Baseline Characteristics | 18 |
| 10.3.1 | Demographics | 18 |
| 10.3.2 | Baseline Characteristics | 18 |
| 10.4 | Surgery Characteristics | 19 |
| 10.5 | Medications for Surgical Procedures, and Prior and Concomitant Medication | s 19 |
| 10.6 | Measurements of Treatment Compliance | 20 |
| 10.7 | Efficacy Analysis | 20 |
| 10.7.1 | Methods of Analysis | 20 |
| 10.7.1.1 | Primary Efficacy Analysis | 20 |
| 10.7.1.2 | Key Secondary Efficacy Analyses | 22 |
| 10.7.1.3 | Secondary Efficacy Analyses | 23 |
| 10.7.1.4 | Exploratory Efficacy Endpoints | 26 |
| 10.8 | Safety Analyses | 28 |
| 10.8.1 | Adverse Events | 28 |
| 10.8.2 | Vital Signs | 30 |
| 10.8.3 | Interim Analysis | 30 |
| 11 | SAMPLE SIZE CALCULATIONS | 30 |
| 12 | REFERENCES | 32 |
| 13 | TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES | 33 |
| 14 | OPIOID RELATED SYMPTOM DISTRESS SCALE (ORSDS) | 36 |
| 15 | LAYOUT OF TABLES, LISTINGS AND FIGURES | 37 |
| 16 | LIST OF TABLES | 39 |
| 17 | LIST OF LISTINGS | 99 |
| 18 | LIST OF FIGURES | 138 |


# 3 LIST OF ABBREVIATIONS

| AE Adverse event ANOVA Analysis of variance ANCOVA Analysis of covariance ATC Anatomical therapeutic class BMI Body mass index bpm Beats per minute CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report d Day |
|---|
| ANCOVA Analysis of covariance ATC Anatomical therapeutic class BMI Body mass index bpm Beats per minute CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| ATC Anatomical therapeutic class BMI Body mass index bpm Beats per minute CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| BMI Body mass index bpm Beats per minute CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| bpm Beats per minute CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| CI Confidence interval CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| CMH Cochran-Mantel-Haenszel CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| CRF Case report form CSE Combined spinal epidural CSR Clinical study report |
| CSE Combined spinal epidural CSR Clinical study report |
| CSR Clinical study report |
| , , |
| d Day |
| d Day |
| ECG Electrocardiogram |
| EMA European Medicines Agency |
| FDA Food and Drug Administration |
| hr, h Hour |
| ICF Informed consent form |
| ICH International Conference on Harmonization |
| ICU Intensive care unit |
| IV Intravenous |
| LOCF Last observation carried forward |
| LS Least square |
| MedDRA Medical dictionary for regulatory affairs |
| MMRM Mixed model repeated measures |
| MPADSS Modified Postanesthesia Discharge Scoring System |
| min Minutes |
| OMED Oral morphine equivalent dose in mg |
| n Number of subjects |
| OR Operating room |
| PACU Postanesthesia care unit |
| PCA Patient-controlled analgesia |
| PO Oral |
| SAE Serious adverse event |
| SAP Statistical analysis plan |
| SD Standard deviation |
| SE Standard error |
| TAP Transversus abdominis plane |
| TEAE Treatment-emergent adverse event |
| TLF Table, listings and figures |
| TUG Timed up-and-go |
| VAS Visual analog scale |
| WHO World Health Organization |
| WHODD World Health Organization – Drug Dictionary |

#### 4 INTRODUCTION

This Statistical Analysis Plan (SAP) describes the planned statistical analysis and reporting of the clinical study 402-C-414 titled "A Multicenter, Randomized, Active-controlled Study to Evaluate the Efficacy and Safety of EXPAREL When Administered via Infiltration into the Transversus Abdominis Plane (TAP) Versus Standard of Care in Subjects Undergoing Elective Cesarean Section."

The structure and content of this SAP provide sufficient detail to meet the requirements identified by the US Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (1999) and the Royal Statistical Society (1993), for statistical practice.

The purposes of this SAP are to:

- Outline the types of analyses and presentations of data that will form the basis for drawing conclusions to the study objectives and hypotheses outlined in the protocol.
- Explain in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices for Good Statistical Practice.

The planned analyses identified in this SAP may be included in the clinical study report (CSR), regulatory submissions, or manuscripts. Post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc, unplanned, or exploratory analyses performed will be clearly identified as such in the final CSR.

The following documents related to clinical study Protocol 402-C-414 were reviewed in preparation of this SAP:

- Original Protocol issued on 16 August 2019.
- Amendment 1 issued on 15Nov2018
- Amendment 2 issued on 07Feb2019
- CRF version 1.0 issued on 04Feb2019
- CRF version 2.0 issued on 05Apr2019
- ICH Guidance on Statistical Principles for Clinical Trials (E9).

The reader of this SAP is encouraged to also read the clinical protocol and other identified documents for details on the planned conduct of this study. Operational aspects related to

collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.

# **5 STUDY OBJECTIVES**

#### 5.1 Primary Objective

The primary objective of this study is to compare total opioid consumption through 72 hours following EXPAREL infiltration into the transversus abdominis plane (TAP) with standard of care (SOC) in subjects undergoing an elective cesarean section (C-section).

#### 5.2 Secondary Objectives

The secondary objectives are to assess efficacy and safety parameters and participant satisfaction.

#### 6 STUDY OVERVIEW

This is a Phase-4, multicenter, randomized, active-controlled study in approximately 182 adult subjects undergoing elective C-section. All subjects will remain in the hospital for up to 72 hours postsurgery.

Subjects will be randomized in a 1:1:1 allocation ratio to receive either:

- Group 1: 150 mcg Duramorph (SOC).
- Group 2: 50 mcg Duramorph + EXPAREL TAP infiltration.
- Group 3: EXPAREL TAP infiltration.

In all treatment groups, a combined spinal epidural (CSE) anesthesia technique may also be used provided the epidural component is not used.

Subjects will be allowed rescue medication upon request to control their pain. Rescue medication will be oral (PO) immediate release oxycodone. If subject cannot tolerate PO medication or fails the PO oxycodone rescue, intravenous (IV) morphine or hydromorphone may be used as rescue medication.

Pain will be assessed using a 10 cm visual analog scale (VAS) for general pain and pain at incision site. Pain will be assessed at multiple prescheduled time points during the study and prior to taking any rescue medication. Subjects will remain in the hospital for up to 72 hours postsurgery.

Other postsurgical assessments include:

- Opioid use
  - Total opioid burden
- Date and time of first unassisted ambulation
- Pain intensity scores using a 10-cm VAS at rest
- Discharge readiness
- Opioid related symptom distress scale
- Date and time of first bowel movement
- Incidence of itching
- Subject's satisfaction with postsurgical pain control
- Calls to physician about pain
- Total time in post-anesthesia care unit (PACU)
- Persistent opioid use at Day 30
- Emergency department (ED) visits
- Recovery from Cesarean Section Scale

#### 7 DEFINITIONS

#### Study Day

If event occurs earlier than the start of study drug, Study Day is calculated as the date of event minus the date of the start of study drug administration. Otherwise Study Day is calculated as the date of event minus the date of the start of study drug administration plus one (+1). Study Day is based on the calendar dates, thus days before the date of surgery have negative values while those on or after the date of surgery are positive.

#### <u>Treatment-emergent Adverse Events</u>

Treatment-emergent adverse events (TEAEs) are the adverse events started on/after the study drug administration.

#### Time 0 (zero)

Time 0 is defined as the date and time of the end of surgery.

#### Time Periods

All scheduled times have a window associated with them (see Time and Events Schedule for individual time point windows). Various time frames are used in the data analyses which are dependent on these windows.

Table 1: Time Window for VAS Assessment

| Defined time VAS Time Point (hrs) | Acceptable Window (hrs) |
|-----------------------------------|-------------------------|
| 12, 24 | ± 1 |
| 48 | ± 2 |
| 72 | ± 4 |

If there are two or more VAS data points that fit into the same time window, the data point close to the center of the window will be used. If two data points are of equal distance to the center, the one with higher VAS score will be used for analysis. For programming purpose, the VAS time point for analysis (ANLO1FL=Y) will be numbered by their schedule, eg, ATPTN = 12, 24, ..., 72. Other VAS time points will be numbered by the VAS time relative to the surgical end time in hours (with 1 decimal point), eg, 47.5.

If after applying the time window, the VAS data point for the scheduled window becomes missing, it will be imputed as per Section 10.1.1.3.

#### Baseline

Baseline is defined as the last available measurement or assessment prior to the start of study treatment.

#### Ready for Discharge

Ready for discharge is defined as a total score of 9 or more on the Modified Postanesthesia Discharge Scoring System (MPADSS). The total score is the sum of all scores. If there are missing data, then the total score will not be calculated.

#### Discharge Time

Discharge time is defined as Discharge day - admission day + 1.

#### Time to Event

Time to event will be calculated as the time from end of surgery to time of event in hours.

#### Opioid-free

Opioid-free is defined as not received opioid rescue medication during the time interval.

#### **Opioid-sparing**

Opioid-sparing is defined as meeting both of the following conditions:

- Total opioid consumption through 72 hours (all doses) ≤15mg (oral morphine equivalent dose [OMED])
- Total itching scores at 12, 24, 48 and 72 hours ≤1;

No opioid-related AEs - Nausea/Abdominal distension/Dizziness

#### 8 ANALYSIS SETS

#### 8.1 Safety set

The safety set will be defined as follows

- Group 1 subjects who underwent C-section surgery and received SOC as scheduled
- Group 2 and Group 3 subjects, who underwent C-section surgery and received study drug through TAP infiltration as scheduled.

All analyses based on the safety set will be by actual treatment received.

#### 8.2 Efficacy set

All the subjects in Safety Set who completed through 72 hours postsurgery. All analyses based on the efficacy set will be by planned treatment at randomization.

#### 8.3 Sensitivity set

All the subjects in Efficacy set who did not receive the correct TAP infiltration based on ultrasound image/video will be excluded from sensitivity analysis. The ultrasound image/video for each patient was reviewed by independent ultrasound review committee. Incorrect TAP infiltration would only be confirmed if two rejections are received.

#### 9 STUDY ENDPOINTS

#### 9.1 Efficacy Endpoints

#### 9.1.1 Primary Efficacy

The primary endpoint is the total opioid consumption (in mg of oral morphine equivalent dose [OMED, see 9.3.1]) to cover postsurgical pain in morphine equivalents through 72 hours. Duramorph, though administered prior to surgery, is used to cover postsurgical pain thus is included in opioid consumption to cover postsurgical pain.

#### 9.1.2 Key Secondary Efficacy

The key secondary endpoint is the average postsurgical itching scores through 72 hours.

#### 9.1.3 Secondary Efficacy

The following secondary endpoints will be analyzed:

Postsurgical itching scores through 12, 24 and 48

- Total Opioid Consumption through 24 and 48 hours, Day 7 (168 hours) and Day 14 (336 hours)
- Average VAS pain intensity scores (general pain and pain at incision site) through 24, 48 and 72 hours after surgery or hospital discharge, whichever occurs first
- Percentage of postsurgical opioid-free and opioid-sparing subjects through 72 hours
- ORSDS at 24, 48, and 72 hours after surgery or at hospital discharge, whichever occurs first
- Proportion of subject discharge-ready at 24, 48, and 72 hours or at hospital discharge, whichever occurs first
- Overall assessment of subject satisfaction with pain control at 72 hours or at hospital discharge, whichever occurs first
- Recovery Cesarean Section Scale

#### 9.1.4 Exploratory Efficacy

- Total postsurgical opioid consumption (in mg of OMED) in morphine equivalents through 72 hours, excluding duramorph administered prior to surgery.
- Length of hospital stay
- Number of unscheduled phone calls or office visits related to pain from discharge through Day 14
- ED visits
- Persistent opioid use at Day 30
- Time spent in the post-anesthesia care unit (PACU)
- Time to first unassisted ambulation.
- Time to first bowel movement

#### 9.2 Safety Endpoints

- Safety will be assessed using the following: Incidence of treatment-emergent AEs (TEAEs) and SAEs through Day 14
- Vital signs at scheduled time points

#### 9.3 Efficacy Assessment

#### 9.3.1 Opioid Dose Conversion

Opioids dose will be converted to oral morphine equivalent dose (OMED mg) using the conversion factor from Table 2 for all summaries. Total opioid dose is the oral morphine


equivalent sum of all opioids taken during the time interval of interest. Subjects with no opioid use during the period in question will be assigned a dose of 0 mg for summaries.

| Table 2. Conversion Factors to IV and Oral Morphine Equivalent Dose from Other Opioids | | | | |
|---|---|---|---|---|
| Medication | Unit | Route | IV Morphine<br>Conversion<br>(Multiplication)<br>Factor | Oral Morphine<br>Conversion<br>(Multiplication)<br>Factor |
| Duramorph | mcg | IT | 0.1 | 0.3 |
| Oxycodone, Oxycocet, Percocet, acetaminophen-oxycodone | mg | РО | 0.5 | 1.5 |
| Morphine | mg | IV, IM, SC | 1 | 3 |
| Morphine | mg | РО | 0.33 | 1 |
| Hydromorphone (Dilaudid) | mg | IV, IM, SC | 6.67 | 20 |
| Hydromorphone (Dilaudid) | mg | РО | 1.3 | 4 |
| Fentanyl | mg | IV, PO, IM | 100 | 300 |
| Hydrocodone combination product - Vicodin,<br>Norco, Lorcet, Lortab, hydrocodone-<br>acetaminophen, Ketobemidone | mg | РО | 0.33 | 1 |
| Codeine combination product - Tylenol 3, acetaminophen-coedine, Paracetamol Forte, Tylenol 4 | mg | PO | 0.05 | 0.15 |
| Ultram, Tramadol, Tramacol hydrochloride | mg | PO, IM | 0.08 | 0.25 |
| Demerol, Meperidine, Pethidine | mg | IV, SC | 0.1 | 0.3 |
| Demerol, Meperidine, Pethidine | mg | РО | 0.033 | 0.1 |
| Ketobemidone, Oxycodone | mg | IV | 1 | 3 |
| Nalbuphine/Nallouphine (Nubain/Manfine) | mg | IV, IM, SC | 1 | 3 |
| PO = oral, IV = intravenous, IM = Intramuscular | , SC = sı | ubcutaneous | , VAS = visual analog | scale. |

# 9.3.2 Average Postsurgical VAS pain Intensity Scores Through 72 Hours or Hospital Discharge, Whichever Occurs First.

To calculate average of postsurgical VAS pain intensity score through 72 hours or hospital discharge, whichever occurs first, we collected pain scores for each subject at each prespecified time. Subjects who did not report any pain score at any time point after surgery will be excluded from this analysis. All the pain scores will be first adjusted for rescue medication if necessary (see 10.1.1.3). Then the remaining missing pain scores will be imputed the median pain score from the patients in the same treatment group and same scheduled time point (see Section 10.1.1.3). The area under the pain-time curve (AUC) is derived using the trapezoidal

rule (see formula below) on the adjusted and imputed pain scores. AUC will start with the first obtained postsurgical pain assessment. All pain assessments through 72 hours after surgery, both scheduled and unscheduled ones, will be included in deriving AUC. Exact assessment times will be used in deriving AUC.

$$AUC = \{\sum (p_i + p_{(i-1)})(t_i + t_{(i-1)})\} / 2$$

where pi is the VAS pain score at time i and  $t_i$  is the time, in hours, from end of surgery. Note  $t_1$  is 12 hours postsurgery. It is the first time VAS score is collected.

The next step is to obtain the average pain score through 72 hours or hospital discharge from AUC. This will be accomplished by dividing AUC by the time interval between first pain assessment and last assessment for the AUC calculation. For example, if the first pain assessment time and the last pain assessment time used to calculate AUC for a subject were 5.6 hours and 72.2 hours respectively, then the average pain score through 72 hours or hospital discharge would be AUC divided by 66.6 (72.2-5.6 = 66.6).

Average postsurgical pain intensity score will be calculated for general pain and pain at incision site.

# 9.3.3 Opioid Related Symptom Distress Scale (ORSDS)

The Opioid-Related Symptom Distress Scale (ORSDS) is a 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 10 symptoms. The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS is the average of 10 symptom-specific scores (see Section 14). The ORSDS has been validated for outpatient laparoscopic cholecystectomy (under general anesthesia) by assessment of internal consistency, content validity, construct validity, principal components analysis, known group validity, responsiveness, and opioid dose dependency.

# 9.3.4 Subject Satisfaction with Pain

The subject's satisfaction with postsurgical pain control will be conducted at 72 hours after surgery (or at hospital discharge, whichever occurs first), and will be assessed using a 5-point Likert scale as follows: 1. Extremely dissatisfied; 2. Dissatisfied; 3. Neither satisfied nor dissatisfied; 4. Satisfied; 5. Extremely satisfied. Sum of the scores will be used for analysis.

#### 9.3.5 Pain Surgical Fear Questionnaire (SFQ)

The SFQ is an eight-item instrument for the assessment of self-reported surgical fear, which can be divided into short-term (SFQ-s) and long-term (SFQ-l) surgery-related fears. All items are scored on an eleven-point numeric rating scale (NRS) ranging from 0 (not at all afraid) to 10 (very afraid). This results in a score of 0-40 for each subscale. Items are: 1. afraid of operation, 2. anesthesia, 3. postoperative pain, 4. Side effects, 5. health deterioration, 6. failed operation, 7. incomplete recovery, 8. long duration of rehabilitation. Sum of the two subscale SFQ scores by treatment group will be used for analysis.

## 9.3.6 Pain Calls to Physician (Single Question)

As part of the phone call to physician on Day 14, the subject will be asked pain related to surgery, and will be assessed using a 4-point Likert scale as follows: 1. 0 (I have not called my doctor); 2. 1-2 times; 3. 3-5 times; 4. More than 5 times.

## 9.3.7 Persistent Opioid Use

As part of the phone call to physician on Day 30, subjects will be asked if they were currently taking opioid for pain and they can either respond as yes or no. Persistent opioid use is defined as those patients who respond yes to the Day 30 opioid use question.

#### 9.3.8 Recovery from Caesarean Section Scale (RCSS)

At 24, 48, and 72 hours postsurgery or hospital discharge, whichever comes first, subjects are asked to rate their answer (1 = strongly disagree and 7 = strongly agree) to each of the 9 RCSS questions.

#### 10 STATISTICAL METHODS OF ANALYSIS

#### 10.1 General Principles

The statistical analyses will be reported using summary tables, listings, and figures (TLFs). All analyses and tabulations will be performed using SAS® Version 9.4 or later. Continuous variables will be summarized using descriptive statistics [sample size (n), mean, standard deviation (SD), minimum, median, and maximum]. Categorical variables will be tabulated with number and percentage of unique subjects. Unless otherwise noted, percentages will be calculated using the number of subjects in the respective treatment group and analysis set as the denominator and presented with only those categories appearing in the data.

Tables will present 150 mcg Duramorph + SOC, 50 mcg Duramorph + EXPAREL and EXPAREL as separate columns.

#### **10.1.1 Handling Missing Values**

#### 10.1.1.1 Total Postsurgery Opioid Consumption

For the calculation of the total postsurgical opioid consumption, both opioid rescue medication before hospital discharge and opioid pain medication in the daily diary after discharge will be included. If opioid is taken on the discharge day but time of dosing is missing, it will be imputed as time of discharge or 12:00 pm on the discharge day, whichever is later. If opioid is taken after the day of discharge and time of dosing is missing, it will be imputed as 12:00 pm the day after discharge.

Study subjects will be given an ePRO device or an app on their smart phone to report pain score and medications they used at home. We expect that all medications will be entered, except when patients discontinued due to AE or death after surgery.

#### 10.1.1.2 Postsurgical Itching Scores through 72 hours

No imputation will be done on the missing itching score. The missing mechanism were assumed missing at random (MAR). Under this assumption the MMRM analysis (see 10.7.1.2.1) is considered unbiased.

#### 10.1.1.3 VAS Pain Intensity Scores

VAS pain intensity scores will first be adjusted by the amount of opioid taken before pain assessment using following method.

- For pain intensity scores on or before the scheduled 24 hours (on or before the exact 24 hours if the scheduled 24 hour pain score is missing), first calculate the total opioid amount (oral morphine equivalent dose, see section 9.3.1.3) that have been taken before this pain assessment (total\_opi). Then the imputed pain score will be the sum of the original pain score and one tenth of the natural logarithm of total\_opi.
- For pain intensity scores after the scheduled 24 hours (after the exact 24 hours if the scheduled 24 hour pain score is missing), first calculate the total opioid amount that have been taken from 24 hours before this pain assessment (total\_opi). Then the imputed pain score will be the sum of the original pain score and one tenth of the natural logarithm of total\_opi.

After adjustment, missing scheduled VAS pain intensity scores will be replaced by the median of non-missing scores from the same scheduled time point and same treatment group.


#### 10.1.1.4 Exposure, Surgery, and Rescue Medication Date or Time

It is expected that all necessary information on study drug exposure, surgery, and postsurgical rescue medication dates and times will be complete. Any such information that is missing and cannot be obtained through query resolution may be imputed, on a case-by-case basis, in a conservative manner that minimizes bias. For example, if pain medication taken on Day 1 has no time of administration recorded, the imputed time will be the end of surgery plus 1 minute.

#### 10.1.1.5 Adverse Event or Concomitant Medications Dates or Times

For AEs with missing or partially missing start date/time, the following imputation rules will be applied for the determination of treatment-emergent status:

For partial start date/time:

- If the year is unknown, then the date will be assigned the date and time of first dose of study treatment.
- If the year is known to be different from the year of the first dose, then missing month and day will be imputed as the first month and first day of the month.
- If the year is known to be the year of the first dose,
  - a) If the month is unknown or is the same as the month of the first dose, then the missing month and day will be imputed by the month and day of the first dose.
  - b) If the month is known to be different from the month of the first dose, then the missing day is imputed as 01 (first day of the month).
- If the time is unknown, then:
  - a) If the date (day, month, and year) matches the date of the administration of study drug, then the time of the study treatment will be used to impute the missing time.
  - b) Otherwise, '00:00' will be assigned.

For medications with missing or partially missing dates, Section 10.5 provides rules for the determination of prior or concomitant status.

#### 10.1.1.6 Adverse Event Severity or Relationship to Study Drug

If severity of an AE is not reported, then for tables of AEs by severity, the event will be classified as 'Severe' and will be footnoted for the table to indicate this imputation. If relationship to study drug is not reported for an AE, then for tables of study-drug related AEs, the event will be assigned the relationship of 'definite'. Tables presenting related AEs will include all AEs with relationships of 'possible', 'probable' or 'definite' as assessed by the investigator.


#### 10.1.1.7 Time to Event

For calculating time to an event when only the hour is reported, the minutes will be set to zero.

#### **10.1.2** By-Center Analyses

By-site summaries will be presented for disposition, demographics, primary efficacy endpoint and secondary efficacy endpoints. In the by-site analysis, analysis stratified by site or adjusted for site as covariate, the small sites will be pooled into one pseudo site. Pseudo site will be numbered as SITEID 999, including SITEID 104,105,108,109,112,116,120,121,122 and 123

#### 10.1.3 Non-Inferiority Margin (NIM)

For VAS pain scores, several studies used 0.8 or 1 as non-inferiority margin. We chose a more conservative NIM of 0.5 which is the same to our previous c-section study named "A Multicenter, Randomized, Double-blinded, Active-controlled Study to Evaluate the Safety and Efficacy of EXPAREL When Administered via Infiltration into the Transversus Abdominis Plane (TAP) Versus Bupivacaine Alone in Subjects Undergoing Elective Cesarean Section".

For postsurgical opioid consumption through 72 hours, from our previous c-section study listed above, postsurgical opioid consumption for bupivacaine group (which is very similar to 150 mcg Duramorph + SOC in this study) is around 30 mg OMED. Some previous studies using opioid consumption as primary endpoint use 30 mg in a 24h interval as non-inferiority margin and previous literature indicate difference of 10.6 mg in IV morphine equivalent dose (31.8 oral morphine equivalent) daily is the clinical different threshold. These difference will be more than 1 on natural logarithm scale for 72 hour interval. To be conservative, we choose 0.8 (on natural logarithm scale) to be our non-inferiority margin (NIM).

#### **10.2 Subject Disposition**

Subject disposition summaries will include the number of subjects

- Screened,
  - Screen failure
  - Enrolled (ie, randomized)
- Randomized
  - o Randomized not treated,
  - Randomized treated.
- In the safety analysis set,
- In the efficacy set,
- In the sensitivity set,
- Completed the study as planned,
- Discontinued from the study, and

Reasons for discontinuation from the study.

Percentages will be reported for the screen failures and enrolled using the number of subjects screened as the denominator; other percentages will use the number of subjects randomized and treated as denominator, unless otherwise noted.

The safety analysis and enrollment data will be presented as treated. All other data will be presented as randomized.

The disposition summary will present the data for each treatment group. This summary table will present overall sites and for each site separately.

#### 10.3 Description of Demographics and Baseline Characteristics

#### 10.3.1 Demographics

The summary of demographic data will present:

- Age (years) descriptive statistics
- Sex n (%)
- Ethnicity n (%)
- Race n (%)
- Country n (%)

Age is calculated from the date the subject signed the informed consent form (ICF) and birth. It is presented as the number of years between, rounding down to the nearest integer year.

The demographic summary will present the data for each treatment group. Summaries will be provided for each (safety and efficacy) analysis set separately.

#### 10.3.2 Baseline Characteristics

The summary of baseline characteristic data will present:

- American Society of Anesthesiologists (ASA) Classification n (%)
- Baseline ECG interpretation
- Height (cm)
- Weight (kg)
- Body Mass Index (BMI) (kg/m²)
- Surgical Fear Questionnaire (SFQ)

Weight in pounds will be converted to kilograms using the conversion factor of 2.2046 pounds to 1 kilogram. Height in inches will be converted to centimeters using the conversion factor of 2.54 centimeters to 1 inch.

Baseline characteristics summaries will present the data for each treatment group. Summaries will be provided for each (safety and efficacy) analysis set separately.

Descriptive statistics (n, mean, SD, median, minimum and maximum) will be provided for continuous variables. The number and percent of subjects will be tabulated for the categorical variables.

#### **10.4 Surgery Characteristics**

Surgery characteristics including type of anesthesia (general, spinal, or other), use of intraoperative medication (yes or no), use of CSE anesthesia (yes or no), administration of the epidural component of the SCE (yes or no), and duration of surgery will be summarized using descriptive statistics. Summaries will be provided for each (safety and efficacy) analysis set.

Duration of surgery is calculated as the difference between the end of surgery and start of surgery times and reported in hours.

#### 10.5 Medications for Surgical Procedures, and Prior and Concomitant Medications

All medications will be coded using the World Health Organization Drug Dictionary (WHODDE Sep 2018) and will be classified according to the anatomical therapeutic chemical classification term (ATC4) and preferred term (PT).

Preoperative, intraoperative, CSE, multimodal pain, postoperative pain, prescription daily pain, and rescue medications are medications given as part of the surgical procedure with start and stop dates on the day of surgery and start and stop times overlapping with the surgery start and stop times.

Prior and Concomitant medications are medications collected on the Prior/Concomitant Medication eCRF page.

Prior medications are defined as medications with a stop date and time prior to the start of study drug administration.

Concomitant medications are defined as medications taken after the start of study drug administration (i.e., started prior to the start of study drug administration and continued after or started after the start of study drug administration).

For the determination of the prior and concomitant status, these rules will be followed for incomplete dates.

- If the medication stop date is partially missing,
  - o If the year and month indicate the stop date is before study drug administration, it is Prior medication.

- Otherwise, it is concomitant medication.
- If the medication stop date is completely missing, it is concomitant medication.

All medications will be summarized separately by category using n (%) of subjects for each treatment group and across treatment groups by ATC3 term and PT for the safety analysis set. Subjects may have more than one medication per ATC3 and PT. At each level of subject summarization, a subject will be counted once if one or more medications are reported by the same subject at that level.

All medications will be included in the data listing.

#### **10.6** Measurements of Treatment Compliance

Study drug is administered by the site personnel, therefore compliance is assured.

## **10.7 Efficacy Analysis**

For Primary and Secondary Efficacy Analyses, descriptive statistics that are appropriate for the efficacy variable will also be shown by site, but no statistical analyses will be performed within a site. All efficacy analyses will be performed on the efficacy analysis set.

#### 10.7.1 Methods of Analysis

For Primary and Secondary Efficacy Analyses, descriptive statistics appropriate for the efficacy variable will be presented overall and by site. No statistical comparison will be made within a site.

# 10.7.1.1 Primary Efficacy Analysis

Total opioid consumption (OMED mg) will be summarized by treatment group for the total dose consumed between 0 and 72 hours after the end of surgery. Presurgery duramorph, used to treat postsurgery pain, is counted in the total opioid dose consumption. For the frequency count of number of subjects receiving opioid medications, subjects will be counted only once regardless of how many times subjects have received the medications. The summary table will include number of subjects receiving postsurgical opioids, geometric mean and coefficient of variation (CV%), median, minimum and maximum.

Tests for the treatment effect will be based on the following one-sided null hypothesis and alternative hypothesis:

 $H_{01}$ : Mean 0-72 hour opioid consumption in EXPAREL group is not different from that in 150 mcg Duramorph (SOC) group.

 H<sub>a1</sub>: Mean 0-72 hour opioid consumption is less in EXPAREL group than in 150 mcg Duramorph (SOC) group.

- H<sub>02</sub>: Mean 0-72 hour opioid consumption in EXPAREL + 50 mcg Duramorph group is not different from that in 150 mcg Duramorph (SOC) group
- H<sub>a2</sub>: Mean 0-72 hour opioid consumption is less in EXPAREL + 50 mcg Duramorph group than in 150 mcg Duramorph (SOC) group.

A one-sided test will be performed at 2.5% level of significance comparing each of the two dose arms of EXPAREL (EXPAREL and EXPAREL + 50 mcg Duramorph) versus 150 mcg Duramorph (SOC).

To test for significant differences between each of the two dose arms of EXPAREL (EXPAREL + 50 mcg Duramorph and EXPAREL) and the 150 mcg Duramorph (SOC), an analysis of covariance (ANCOVA) model with treatment and site as the main effects, age and height as covariates will be applied to the natural log-transformed total dose. If a subject never received an opioid medication, the total dose will be assigned 3.75 mg OMED prior to the log-transformation. The LS means of the two doses of EXPAREL (EXPAREL + 50 mcg Duramorph and EXPAREL) and 150 mcg Duramorph (SOC), LS mean difference (EXPAREL + 50 mcg Duramorph minus 150 mcg Duramorph (SOC)and EXPARE minus 150 mcg Duramorph (SOC)), two-sided 95% CI for the LS mean difference, and the one-sided p-value will be reported after back transformation (ie, taking exponential) to the original OMED scale.

In addition to the presentation for the between group difference, the percent reduction in total OMED will also be presented. The % reduction is derived as follows,

% Reduction=100% x {LSM\*<sub>150</sub> mcg Duramorph(SOC) - LSM\*<sub>EXPAREL+50mcg</sub> Duramorph }/LSM\*<sub>150</sub> mcg Duramorph(SOC)

where LSM\* is back-transformed least square mean estimate from the ANCOVA.

The primary analysis for the primary endpoint is based on the Efficacy evaluable population.

#### 10.7.1.1.1 Multiplicity Adjustments

For the efficacy analyses, pairwise comparison of the active dose groups (EXPAREL+50 mcg Duramorph and EXPAREL) will be compared to 150 mcg Duramorph (SOC) following spinal anesthesia using the 1-sided 0.025 alpha level for the efficacy analysis set.

To control the family-wise error rate at one-sided 2.5% significance level, a fixed sequence procedure (Westfall et al 1999) will be performed to test the ordered null hypotheses below at 2.5% significance level.

1)  $H_{01}$ : Mean 0-72 hour opioid consumption in EXPAREL group is not different from that in 150 mcg Duramorph (SOC) group.

2)  $H_{02}$ : Mean 0-72 hour opioid consumption in EXPAREL group is not different from that in 150 mcg Duramorph (SOC) group.

First,  $H_{01}$  will be tested at 2.5% significance level for the primary endpoint. If  $H_{01}$  is rejected, it will be claimed that the EXPAREL is superior to 150 mcg Duramorph (SOC), then  $H_{02}$  will be tested at 2.5% significance level. If  $H_{02}$  is rejected, then it will be concluded that both EXPAREL and EXPAREL + 50 mcg Duramorph groups are superior to 150 mcg Duramorph (SOC) group. If  $H_{01}$  is not rejected, then  $H_{02}$  will not be tested and the conclusion will be that neither treatment groups are efficacious.

#### 10.7.1.1.2 Subgroup Analysis of Primary Efficacy Endpoint

The analysis of the primary endpoint will be repeated for selected subgroups such as

- Age (<35, and ≥35),</li>
- Race (White and Non-White),
- BMI (<25, 25 to <30, and ≥30+ kg/m²)</li>
- Number of prior C-sections (0, 1+),
- Discharge Time (Discharged on or before Day 3, Discharged on or after Day 4), and
- Subjects with or without anxiety medical history.

Note because of the small sample sizes, all subgroup analysis will be performed without adjusting/stratifying by site

#### 10.7.1.2 Key Secondary Efficacy Analyses

#### 10.7.1.1.1 Average Postsurgical Itching Scores Through 72 Hours

Postsurgical itching scores (at PACU, 12, 24, 48, and 72 hrs) will be analyzed using an MMRM model with treatment group, site, visit and treatment-by-visit interaction as main effect, age and height as covariates. LS means of each treatment group, LS mean differences between each pair of treatment groups and p-value of each LS mean differences will be presented. The average itching score through 72 hours is estimated by the LS grand mean.

A sample SAS code is provided as follows.

```
PROC MIXED DATA=XXXX;

CLASS trtp usubjid visit siteid;

MODEL Response = siteid age height trtp visit trtp*visit / DDFM=kr2;

REPEATED visit / SUBJECT=usubjid(trtp) TYPE=UN;

LSMEAN trtp*visit/ PDIFF ALPHA=0.05;

LSMEAN trtp / PDIFF;
```

Note: usubjid is subject ID, trtp is treatment variable, visit is the nominal study visit, and Response is the itching score at the scheduled time point. Depending on the convergence status in the computation, unstructured (UN), Toeplitz (TOEP), 1st order autoregressive [AR(1)] and compound symmetry variance-covariance (CS) matrix will be tried in the order. The final analysis will be based on the first matrix leading to the convergence in the computation.

# 10.7.1.3 Secondary Efficacy Analyses

10.7.1.3.1 Average Postsurgical Itching Scores Through 12, 24, 48 and 72 Hours

These endpoints will be analyzed using the same MMRM approach described in Section 10.7.1.2. Between-group simple contrast at each visit will be derived the ESTIMATE statement.

10.7.1.1.2 Total Opioid Consumption Through 24 and 48 Hours, Day 7 (168 hours) and Day 14 (336 hours)

Each individual timepoint will be analyzed using the ANCOVA model similar to Section 10.7.1.1. Between-group simple contrast will be derived from the LSMEAN statement.

10.7.1.3.3 Average VAS Pain Intensity Scores Through 72 Hours After Surgery or Hospital Discharge Whichever Occurs First

Average VAS pain intensities (general pain and pain at incision site) from 0 to 72 hours or hospital discharge whichever comes first will be derived for each subject as described in Section 9.3.2. They will be analyzed using ANCOVA with treatment and site as main effects, age and height as covariates. Based on the model, the LS Mean and SE will be reported for each treatment group. Non-inferiority and superiority sequential hypothesis testing will be performed afterwards, comparing each of the two dose arms of EXPAREL (EXPAREL + 50 mcg Duramorph and EXPAREL) versus 150 mcg Duramorph (SOC) simultaneously: (1) EXPAREL + 50 mcg duramorph vs. 150 mcg duramorph (SOC), and (2) EXPAREL vs. 150 mcg duramorph (SOC). LS Mean difference and 95% CI will be reported for each comparison.

The testing procedure is the same for each comparison. Here we use (1) EXPAREL + 50 mcg duramorph vs. 150 mcg duramorph (SOC) as an example:

# Hypothesis 1 (non-inferiority):

- H1<sub>o1</sub>: EXPAREL group is inferior to 150 mcg Duramorph (SOC) group with respect to average VAS score.
- H1<sub>a1</sub>: EXPAREL group is not inferior to 150 mcg Duramorph (SOC) group with respect to average VAS score.

# Hypothesis 2 (superiority):

- H2<sub>o1</sub>: EXPAREL group is not superior to 150 mcg Duramorph (SOC) group with respect to average VAS score.
- H2<sub>a1</sub>: EXPAREL group is superior to 150 mcg Duramorph (SOC) group with respect to average VAS score.

To test the two null hypotheses, a stepdown approach will be used by inspecting the 95% confidence interval for group difference as follows:

- Non-inferiority Test for Hypothesis 1.
  - o If the upper bound of the 2-sided 95% confidence interval for the LSM for the difference of average VAS score under  $H1_{o1}$  versus  $H1_{a1}$  is > NIM, then stop the hypothesis tests and declare that the non-inferiority result is not achieved. NIM (non-inferiority margin) = 0.5.
  - o If the upper bound of the 2-sided 95% CI is ≤ NIM then declare that the non-inferiority of EXPAREL+50 mcg Duramorph to 150 mcg Duramorph (SOC) is achieved. Move on to test for H2<sub>01</sub>.
- Superiority Test for Hypothesis 2
  - O If the upper bound of the 2-sided 95% CI is ≥0 for the comparison (EXPAREL+50 mcg Duramorph versus 150 mcg Duramorph (SOC)), then stop the test and declare that the superiority is not achieved for H2<sub>01</sub>.
  - If the upper bound is <0 then declare that the superiority of EXPAREL+50 mcg</li>
     Duramorph to 150 mcg Duramorph (SOC)is achieved.

In the table presentation for the between group comparison, if the superiority test passes, only the 1-sided superiority test p-value will be displayed. If the superiority test fails, only the 1-sided non-inferiority test p-value will be displayed. Margin used for noninferiority test will be 0.5.

Summary and analysis of (general and at incision site) average VAS pain intensity scores through 24, and 48 hours will also be reported.

10.7.1.3.4Percentage of Postsurgical Opioid-Free and Opioid-Sparing Subjects Through 72
Hours

The percentage of opioid-free subjects through 72 hours and hospital discharge will be analyzed using the logistic regression model with treatment, site, age, and height as explanatory variables. Percentage of opioid-free subjects from the model, odds ratios (EXPAREL+50 mcg Duramorph) / 150 mcg Duramorph (SOC) and EXPAREL / 150 mcg Duramorph (SOC), and 95% CI for the odds ratios and p-values will be presented.

Percentage of opioid sparing subjects will be analyzed using the same approach described for percentage of opioid free subjects.

#### Pseudo-code for logistic regression method:

```
ods output OddsRatios=or /* ODDS RATIO AND 95% CL*/
    Diffs=diff(keep=probz) /* 1-SIDED P-VALUE */
    LSMeans=lsm(keep=trtpn mu) /* PROB OF YES */;
proc logistic data=ef1 plots=none;
    class siteid trtpn / param=glm;
    model avalc(event="Yes")=trtpn siteid age heightbl;
    lsmeans trtpn / pdiff=controll('2') ilink;
run;
```

10.7.1.3.5 Opioid Related Symptom Distress Scale (ORSDS) at 24, 48, and 72 Hours After Surgery or at Hospital Discharge, Whichever Occurs First

The ORSDS composite score as well as the 10 symptom-specific ORSDS scores will be summarized by treatment at each assessment time points of 24, 48, and 72 hours after surgery or at hospital discharge, whichever occurs first. Additionally, the ORSDS composite and each of the symptom-specific distress scores will be analyzed using a Mixed-Effect Model for Repeated Measures (MMRM). The model includes treatment, visit, and interaction between treatment and visit as fixed factors. The model parameters will be estimated using restricted maximum likelihood method with unstructured variance-covariance matrix and Kenward-Roger approximation to estimate denominator degrees of freedom. The between-group comparison will be performed using the simple contrast at the respective visits. The LSM of 150 mcg Duramorph (SOC), EXPAREL + 50 mcg Duramorph and EXPAREL, the difference in the LSM (EXPAREL + 50 mcg Duramorph minus 150 mcg Duramorph (SOC) and EXPAREL minus 150 mcg Duramorph (SOC), and 95% CI for the LSM difference will be calculated. Analysis will be performed at 24, 48 and 72 hours.

A sample SAS code is provided as follows.

```
PROC MIXED DATA=XXXX;
```

```
CLASS trtp usubjid visit;

MODEL Response = siteid trtp visit trtp*visit / DDFM=kr2;

REPEATED visit / SUBJECT=usubjid(trtp) TYPE=UN;

Lsmeans trtp*visit/Pdiff alpha=0.05;

RUN;
```

Note: usubjid is subject ID, trtp is treatment variable, visit is the nominal study visit, and Response is respective endpoints. Depending on the convergence status in the computation, unstructured (UN), Toeplitz (TOEP), 1<sup>st</sup> order autoregressive [AR(1)] and compound symmetry variance-covariance (CS) matrix will be tried in the order. The final analysis will be based on the first matrix leading to the convergence in the computation.

10.7.1.3.6Proportion of Subjects Discharge-Ready at 24, 48, and 72 Hours or at Hospital Discharge, Whichever Occurs First

Proportion of subject discharge-ready at each timepoint of 24, 48, and 72 hours or at hospital discharge, whichever occurs first will be analyzed using logistic regression similar to section 10.7.1.3.4

10.7.1.3.70verall Assessment of Subject Satisfaction with Pain Control at 72 Hours or at Hospital Discharge, Whichever Occurs First

Overall assessment of subject satisfaction with pain control at 72 hours or at hospital discharge, whichever occurs first (obtained using a 5-point Likert scale) will be summarized with mean and SD and tabulated with n (%) by treatment group. The between group comparison will be carried out using the using the Cochran-Mantel-Haenszel (CMH) test for row mean score difference (RMS) with modified ridit score.

#### Pseudo-code for CMH method:

```
PROC FREQ;
```

TABLE siteid\*trt\*Y / cmh SCORES=modridit scorout;

RUN;

where, Y is subject satisfaction scores

10.7.1.3.8Recovery from Caesarean Section Scale (RCSS)

Subject rating on each of the 9 scales will be summarized descriptively by treatment group at 24, 48, and 72 hours, or at hospital discharge, whichever occurs first.

- 10.7.1.4 Exploratory Efficacy Endpoints
- 10.7.1.1.1 Total Postsurgical Opioid Consumption (mg) in Morphine Equivalents Through 72 Hours

Total postsurgical opioid consumption (mg) in morphine equivalents through 72 hours or hospital discharge will be analyzed using ANCOVA similar to section 10.7.1.3.3. Non-inferiority comparison will be conducted by comparing the upper bound of the 95% CI for the between treatment difference (in the log-transformed scale) against the noninferiority margin (NIM=0.8). If a subject never received any postsurgical opioid medication, the total dose will be assigned 3.75 mg OMED (half of one oral oxycodone dose) prior to the log-transformation.

# 10.7.1.4.2 Length of Hospital Stay

Length of hospital stay, defined as the surgical facility discharge date/time minus the facility admission date/time, will be summarized descriptively by treatment group.

# 10.7.1.4.3 Number of Unscheduled Phone Calls or Office Visits Related to Pain from Discharge Through Day 14

The number of unscheduled pain-related phone calls per subject after discharge through postsurgical Day 14 will be summarized with mean and SD and tabulated with n (%) of subjects with 0, 1, 2, 3, etc. phone call by treatment.

## 10.7.1.4.4Number of Emergency Department (ED) Visits

The number of ED visits per subject after discharge will be summarized with mean and SD and tabulated with n (%) of subjects with 0, 1, 2, 3, etc. ED visits by treatment.

#### 10.7.1.4.5 Persistent Opioid Use at Day 30

The number (and %) of subjects with persistent opioid use at day 30 after discharge will be summarized by treatment group.

#### 10.7.1.3.6Time Spent in the Post-Anesthesia Care Unit (PACU)

The time spent (hours) in PACU is defined as date/time of admission to PACU minus date/time of discharge from PACU. This endpoint will be analyzed by treatment group using ANCOVA similar to Section 10.7.1.1 Baseline value will be included in the model as covariate and assuming gamma (or normal) distribution and log link function

#### 10.7.1.3.7Time to First Unassisted Ambulation

Time to first unassisted ambulation will be computed in hours as the date and time of the first unassisted ambulation minus the date and time of the end of surgery. If a subject is not administered an ambulation, the time to first unassisted ambulation will be censored at 72 hours after surgery or at the time of last follow-up, whichever is early.

Time to first unassisted ambulation will be analyzed in two steps: Kaplan-Meier Curves for each treatment group with log-rank test for the between group difference. Cox proportional hazards regression with treatment and site as factors, age and height as covariates, followed by chi-squared test. The n (%) of subjects with unassisted ambulation as well as the n (%) of subjects without unassisted ambulation will be presented for each treatment group.

#### 10.7.1.4.8Time to First Bowel Movement

Time to first bowel movement will be computed in hours as the date and time of the first bowel movement minus the date and time of the end of surgery. If a subject does not have bowel movement, the time to first bowel movement will be censored at 72 hours after surgery or at the time of last follow-up, whichever is early. Time to first bowel movement will be analyzed by the method similar to time to first unassisted ambulation.

#### **10.8 Safety Analyses**

Safety assessments in this study consist of adverse events (AEs) and vital signs (VS).

#### 10.8.1 Adverse Events

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA v21.1).

An AE will be considered TEAE if it starts on/after the start time of the first study medication subject received. Specifically, if subjects receive study medications according to the protocol, Group 1 and 2 subjects will use Duramorph and Group 3 subjects will use EXPAREL start time for reference.

If an AE has a partial onset date and time the imputed start dates and time will be used to determine treatment-emergence (Section 10.1.1.5). All AE summaries will present TEAEs only. AEs that are not treatment-emergent will be included in listings but not summarized.

AEs will be summarized using subject incidence table. An overview of TEAE will be presented. This table will include n (%) of subjects with

- Any TEAE
  - Maximum severity: Mild
  - Maximum severity: Moderate
  - Maximum severity: Severe
- At least one related TEAE
- At least one serious TEAE
- Subjects discontinued due to a TEAE
- Died on study

Additionally, n (%) are calculated based on the number of unique subjects within each MedDRA category (eg, preferred term) by treatment group. A subject reporting multiple events of the same category will be counted only once for that category. For summary purpose, AE relationship to the study drug will be grouped into "Unrelated" for "unrelated" or "unlikely related" and "Related" for "possibly", "probably", or "definitely related". For subjects with more than one event coded to the same PT, the subjects will be counted for the categories with the strongest relationship and the greatest severity. The following subject incidence tables will be presented.

- TEAEs by PT (Preferred Term) sorted by the decreasing order of subject incidence in the combined group
- TEAEs by SOC (System Organ Class) and PT sorted alphabetically
- TEAEs by study drug-relationship by SOC and PT
- TEAEs by severity and by SOC and PT
- TEAE of special interest (TEAESI) by SOC and PT

A subject data listing will be provided for all adverse events. Included in the listing are the reported term, PT, SOC, TEAE flag, study day when AE starts, duration, relationship, severity, action taken, outcome, and seriousness category.

Separate data listings will be provided for subjects who die on study, experience SAEs, have TEAEs leading to study discontinuation, or AEs of special interest.

AE of special interest will be extracted based on the MedDRA terms below.

**Table 3. Adverse Events of Special Interest** 

| Group | MedDRA System Organ Class | MedDRA Preferred Terms |
|---|---|---|
| FALL | Injury, poisoning and procedural complications | Fall |
| | Cardiac Disorders | Arrhythmia |
| | Cardiac Disorders | Atrial Fibrillation |
| | Cardiac Disorders | Atrial Tachycardia |
| | Cardiac Disorders | Atrioventricular Block |
| | Cardiac Disorders | Atrioventricular Block First Degree |
| LAST | Cardiac Disorders | Bradycardia |
| LAST | Cardiac Disorders | Bundle Branch Block Left |
| | Cardiac Disorders | Bundle Branch Block Right |
| | Cardiac Disorders | Cardiac Arrest |
| | Cardiac Disorders | Cardiac Failure Acute |
| | Cardiac Disorders | Cardiac Failure Congestive |
| | Cardiac Disorders | Conduction Disorder |


| Group | MedDRA System Organ Class | MedDRA Preferred Terms |
|-------|---------------------------|----------------------------------|
| | Cardiac Disorders | Myocardial Infarction |
| | Cardiac Disorders | Sinus Arrest |
| | Cardiac Disorders | Sinus Arrhythmia |
| | Cardiac Disorders | Sinus Bradycardia |
| | Cardiac Disorders | Sinus Tachycardia |
| | Cardiac Disorders | Supraventricular Tachyarrhythmia |
| | Cardiac Disorders | Supraventricular Tachycardia |
| | Cardiac Disorders | Tachyarrhythmia |
| | Cardiac Disorders | Tachycardia |
| | Cardiac Disorders | Ventricular Extrasystoles |
| | Cardiac Disorders | Ventricular Tachycardia |
| | Nervous System | Dizziness |
| | Nervous System | Dysgeusia |
| | Nervous System | Somnolence |
| | Nervous System | Tremors |

A listing of the mapping of the system organ class and preferred terms to verbatim terms will be presented.

## 10.8.2 Vital Signs

Vitals signs are resting heart rate (bpm), systolic blood pressure (mmHg), and diastolic blood pressure (mmHg). Vital signs will be summarized by treatment group at each assessment time point. Summaries will present both actual and change-from-baseline results.

#### 10.8.3 Interim Analysis

After approximately 20 subjects per treatment group were randomized and treated (i.e., a total of 60 subjects were treated in this study), a preplanned interim analysis was conducted in accordance with Amendments 1 & 2 of the study protocol and the 26Sep2019 Interim Analysis Plan. The decision from the interim analysis was made to enroll a total of at least 140 treated subjects.

# 11 SAMPLE SIZE CALCULATIONS

Assuming a log-normal distribution for total opioid consumption with a 70% coefficient of variation (CV), 5% alpha, an equal randomization ratio, and 80% power, a total of 77 subjects per treatment group will be sufficient to detect a 25% reduction in total opioid consumption. Assuming 5% of the subjects are not evaluable and one of the two EXPAREL groups will be dropped after interim analysis when a total of 60 subjects are treated, a total sample size of

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-414 (C-section TAP) Statistical Analysis Plan

approximately 182 treated subjects is needed. This sample size will be re-evaluated after the interim analysis.

402-C-414 (C-section TAP) Statistical Analysis Plan

#### 12 REFERENCES

Newcombe, RG, Interval Estimation for the Difference between Independent Proportions: Comparison of Eleven Methods. Statist. Med. 17, 873-890 (1998).

Nieto, FJ and J Coresh. Adjusting Survival Curves for Confounders: A Review and a New Method. American Journal of Epidemiology. 1996. Vol. 143, No. 10.

Rubin, DB. (1987). Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons.

Quale, M, G Cunningham, C Foster, and J Hutchins. Addition of transversus abdominis plane infiltration with liposomal bupivacaine to intrathecal morphine for postoperative analgesia after Caesarean delivery: a retrospective study. Abstract 1497. American Society of Regional Anesthesia and Pain Management. 41st Annual Regional Anesthesiology and Acute Pain Medicine Meeting. 31-Mar-2016 to 02-Apr-2016. New Orleans, LA, US.

Saville, BR, JT Connor, GD Ayers, J Alvarez. The Utility of Bayesian Predictive Probabilities for Interim

Monitoring of Clinical Trials. Clinical Trials. May 2014, p485-493, Vol. 11, No. 4.

Schafer, JL. (1997). Analysis of Incomplete Multivariate Data. New York: Chapman & Hall.

# 13 TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES

Please see the Protocol for the full "Time and Events Schedule of Study Procedures".

Table 1. Assessment Schedule (Screening through 72 hours after Surgery)

| Natural Control of the Control of th | Within 30 days | Screening | Ç. | Day 1 | 9 11 11 1 | Hours after Surgery | | |
|---|---|---|---|---|---|---|---|---|
| Study Procedure | of scheduled<br>surgery | (up to 30 days prior<br>to day of surgery) | OR | PACU | 12 hr<br>(± 1hr) | 24 hr<br>(± 1hr) | 48 hr<br>(± 2hr) | 72 hr<br>(± 4hr) |
| Explain study purpose and procedures; obtain signed ICF | $\mathbf{X}^{1}$ | X <sup>1</sup> | | | | | | 61 100 |
| Assess/confirm eligibility | | X | X | | | | | |
| Record/confirm medical and surgical history | | X | X | | | | | |
| Record prior and concomitant medications | K- | X | X | | | | | |
| Record demographics and baseline characteristics | 2 | X | 8 | 8 8 | | | | |
| Measure vital signs (blood pressure, heart rate, respiratory rate, and temperature) | | X <sup>2</sup> | X | $X^{l1}$ | | X | X | X <sup>3</sup> |
| Measure pulse oximetry per SOC10 | | | <b>←</b> | | | $\rightarrow$ | | |
| Physical examination (according to the investigational site's SOC) | | х | X | | | | | |
| Drug screen/alcohol test | | X | | 9 9 | | | | |
| Clinical laboratory tests (hematology and chemistry;<br>Appendix 5) <sup>4</sup> | | х | | | | | | |
| 12-lead electrocardiogram | | X | | | | | | |
| Explain ePRO device and expectations of the subject regarding the device | | X | | | | | | |
| Randomize subject and prepare study drug | | | X | | | | | |
| Administer intrathecal preservative-free morphine injection in conjunction with single-shot spinal anesthesia per the treatment group (Section 13.4) | | | x | | | | | |
| Record surgery start and stop times | | | X | | | | | |
| Perform TAP needle placement and saline hydrodissection under<br>ultrasound guidance using up to 10 mL normal saline (per the<br>treatment group) | | | | x | | | | |
| Capture ultrasound image or video of the TAP needle placement after saline hydrodissection | | | | X | | | | |
| Perform 2-point classic TAP infiltration no more than 90 min<br>after skin-incision closure of the C-section (per the treatment<br>group) | | | | X | | | | |
| Take ultrasound image of the 2-point classic TAP needle<br>placement after study drug infiltration | | | | X | | | | |
| Record start and stop times of study drug infiltration | 9 | | | X | | | | |
| Record intraoperative opioid medications administered and doses | | 6 | X | | | | | |

| | Within 30 days | Screening | | Day 1 | | Hours after Surgery | | |
|---|---|---|---|---|---|---|---|---|
| Study Procedure | of scheduled<br>surgery | (up to 30 days prior<br>to day of surgery) | OR | | 12 hr<br>(± 1hr) | 24 hr<br>(± 1hr) | 48 hr<br>(± 2hr) | 72 hr<br>(± 4hr) |
| Record date, time in and out of the PACU | 1 | | | X | | 2 33 | (2) | |
| Record SFQ (Appendix 6) | | X | | 0. | 50 | a (8 | 307 | |
| Record scheduled 10 cm VAS pain intensity scores (General<br>and Site of Incision) at rest through ePRO <sup>5,6,7</sup> (Appendix 1) | | | | | X | X | X | X |
| Record 10 cm VAS pain intensity (through ePRO) immediately<br>prior to any postsurgical opioid medication administered<br>while in the hospital (Appendix 1) | | | | X | X | X | X | X |
| Record date, time, and dose of all postsurgical pain medication <sup>8</sup> | ( ) | | | X | X | X | X | X |
| Record date, time, and dose of all standardized multimodal pain<br>medications administered | | | | X | X | X | X | X |
| Record date and time of first unassisted ambulation | | | | X | X | X | X | X |
| Record date and time of first bowel movement | | | | X | X | X | X | X |
| Assess itching (Numeric Rating Scale of 0 to 10) | | X | | X11 | X | X | X | X |
| Record overall rating of subject's satisfaction with postsurgical<br>pain control through ePRO (Appendix 3) | | | | | | | 3.71 | X <sup>3</sup> |
| Record RCSS through ePRO (Appendix 4) | | | | 8 | | X | X | $X^3$ |
| Record ORSDS through ePRO (Appendix 7) | | | | 8 | | X | X | X |
| Assess discharge readiness <sup>9</sup> (Appendix 2) | | | | G. | 50 | X | X | X |
| Record concomitant medications for treatment of AEs | | X | X | X | X | X | X | X |
| Record AEs/SAEs (starting at signing of ICF) | | X | X | X | X | X | X | X |

- Potential participants may provide informed consent up to 30 days before their scheduled surgery. If a subject can only be screened on the day of surgery, the consent process
  must be started at least 24 hours prior to the day of surgery in order to ensure ample time for the subject to review the ICF and have all her questions answered by the
  investigator/study staff prior to providing informed consent. Screening procedures that are SOC at the institution may be completed prior to written informed consent. Any
  screening procedures that are not SOC, must be completed after written informed consent is provided and prior to surgery.
   If a subject can only be screened on the day of surgery, the informed consent process must still be started at least 24 hours prior to the conduct of any screening procedures
  that are not considered SOC at the institution and such procedures may not be performed until written informed consent is provided.
- 2. Vital signs at screening will include height, weight, blood pressure, heart rate, respiratory rate, and temperature.
- 3. At 72 hours postsurgery or prior to hospital discharge, whichever occurs first.
- Clinical laboratory tests will be conducted in accordance with the investigator's SOC, including direct bilirubin; either gamma-glutamyl transpeptidase and lactate dehydrogenase or alanine transaminase and aspartate transaminase; and either serum creatinine or blood urea nitrogen.
- To assess pain intensity (VAS) general and at incision site at rest, the subject should rest quietly in a supine or seated position that does not exacerbate her postsurgical pain for 3-5 minutes before entering the pain score. This assessment should not be completed immediately following assessment of ambulation.
- 6. If a subject is discharged prior to any of the scheduled VAS assessments (general and at incision site) to be collected at 12 to 72 hours after surgery, a member of the study site staff will contact the subject at the appropriate scheduled times (i.e., the time of each assessment scheduled to be collected that occurs after hospital discharge) to remind her to complete the VAS and ORSDS assessments and to record the scheduled assessments in the device. This will ensure that, for any subject discharged prior to 72 hours, all VAS and ORSDS assessments required for calculation of the study endpoints are captured. These phone calls will only be made if a subject is discharged prior to 72 hours.

Pacira Pharmaceuticals, Inc. EXPAREL

402-C-414 (C-section TAP) Statistical Analysis Plan

- 7. For pain intensity scores at 12, 24, 48, or 72 hours, if the subject is sleeping, do not wake her to assess pain. If she awakens within the assessment window (i.e., 1 hour for the 12- and 24-hour assessments, 2 hours for the 48-hour assessments, and 4 hours for the 72-hour assessments), a pain score may be collected then.
- 8. Subjects should only receive opioid pain medication (e.g., morphine, hydromorphone [Dilaudid], oxycodone) upon request for breakthrough pain.
- 9. Discharge readiness will be assessed at 24, 48, and 72 hours, or hospital discharge, or until the subject attains score of 9, whichever occurs first.
- 10. Pulse oximetry measured once prior to surgery and per your site's SOC from surgery end up to 24 hours.
- 11. Assess vital signs (blood pressure, heart rate, respiratory rate, and temperature) and itching in PACU prior to PACU discharge.

Note: No more than 30 days should pass between signing of the ICF and performance of the surgery. Screening on the day of surgery will be permitted but is discouraged.

Note: The end of surgery is defined as the time of skin-incision closure of the C-section wound (following delivery and prior to TAP infiltration).

AE=adverse event; C-section=cesarean section; ePRO=electronic patient-reported outcome; hr=hour(s); ICF=informed consent form; OR=operating room; ORSDS=Opioid Related Symptom Distress scale; PACU=post-anesthesia care unit; RCSS=Recovery from Cesarean Section scale; SAE=serious adverse event; SFQ=Surgical Fear Questionnaire; SOC=standard of care; TAP= transversus abdominis plane; VAS=visual analog scale

# 14 OPIOID RELATED SYMPTOM DISTRESS SCALE (ORSDS)

| Symptoms | Did not<br>have | (If yes), how often did<br>you have it? | | | | (If yes), how severe was it usually? | | | | (If yes), how much did it distress<br>or bother you? | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| | | Rarely | Occasionally | Frequently | Almost Constantly | Slight | Moderate | Severe | Very Severe | Not at all | A little Bit | Somewhat | Quite a Bit | Very Much |
| Fatigue | | | | | | | | | | | | | | |
| Drowsiness | | | | | | | | | | | | | | |
| Inability to concentrate | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | |
| Dizziness | | | | | | | | | | | | | | 9 |
| Constipation | | | | | | | | | | | | | | |
| Itching | | | | | | | | | | | | | | |
| Difficulty with urination | | | | | | | | | | | | | | |
| Confusion | | | | | | | | | | | | | | |
| Retching/vomiting | | | # of | episodes | | | | | | | | | | |
## 15 LAYOUT OF TABLES, LISTINGS AND FIGURES

The following are planned summary tables. Tables will be numbered according to the nomenclature used to support the CSR. The final table numbering may be different from the SAP. No amendment will be made for changes in table numbering. All headers, titles, footnotes, and footers specified in the table mock-ups will be displayed in the produced output unless otherwise specified. Notes to programmers will not be included in the tables.

Tables and listings will have 10-point font size. Listings font size may be reduced to 9 point if needed. The TLFs will have either Times New Roman, Courier New or SAS Monospace type face. All final TLFs will be provided in both PDF and Word (or RTF) file formats.

Percentages should not appear if the count is zero.

Italicized text in the TLF mock-ups indicate notes to programmers and is not to appear on any TLF.

Note headers and footers on mock-ups are reflective of the SAP document and are not intended to appear on the TLFs.

Titles on the TLFs in the mock-ups are presented left-justified as a single line of text. However, the presentation for final TFLs should be center-justified with the TLF number on one line and the remaining titles on multiple lines of text where the line breaks are delimited by hyphens (-) in the TLF mock-ups titles. For example, for Table 14.2-1.1a the title in the mock-up appears as:

Table 14.2-1.1a: Analysis of Postsurgical Total Opioid Consumption (OMED mg) Through 72 hours - Efficacy Analysis Set

but should appear as follows on the final TLF:

Table 14.2-1.1a

Analysis of Postsurgical Total Opioid Consumption (OMED mg) through 72 hours Efficacy Analysis Set

The title format in the mock-ups is due to limitations of MS Word. The mock-up format enables MSWord to generate a table of contents for the mock-ups.

For categorical variables, if subjects have missing values (example Race), a "missing" category will be added as appropriate.

All tables will present treatment Active (for EXPAREL+50 mcg Duramorph or EXPAREL) and 150 mcg Duramorph (SOC) as separate columns.

On all figures, EXPAREL+50 mcg Duramorph will be represented in red with solid lines and dots, EXPAREL will be represented in blue with solid lines and filled squares and 150 mcg Duramorph (SOC) will be represented in black with solid lines and filled diamonds.

On all listings the treatments, in the order of appearance, are: EXPAREL+50 mcg Duramorph, EXPAREL, 150 mcg Duramorph (SOC)and, if applicable, NOT RANDOMIZED. Always insert a page break between treatments.

On all listings sort within treatment by site, subject, with further sorts dependent on listing.

The shell provides a general guidance for how the data will be presented. The actual presentation may be modified to accommodate the page size restriction.

For TFLs with multiple pages, page numbers will be included.

All TFLs will have SAS program names and folder names and date/time stamp in the footnote for tracking purpose.

| 16 LIST OF TABLES | |
|---|---|
| TABLE 14.1-1: SUMMARY OF SUBJECT DISPOSITION – ALL SCREENED SUBJECTS | 43 |
| TABLE 14.1-2.1: SUMMARY OF SUBJECT DEMOGRAPHICS – EFFICACY ANALYSIS SET | 45 |
| TABLE 14.1-2.2: SUMMARY OF SUBJECT DEMOGRAPHICS – SENSITIVITY ANALYSIS SET | 46 |
| TABLE 14.1-2.3: SUMMARY OF SUBJECT DEMOGRAPHICS – SAFETY ANALYSIS SET | 46 |
| TABLE 14.1-3.1: SUMMARY OF SUBJECT BASELINE CHARACTERISTICS – EFFICACY ANALYSIS SET | 47 |
| TABLE 14.1-3.2: SUMMARY OF SUBJECT BASELINE CHARACTERISTICS – SENSITIVITY ANALYSIS SET | 49 |
| TABLE 14.1-3.3: SUMMARY OF SUBJECT BASELINE CHARACTERISTICS – SAFETY ANALYSIS SET | 49 |
| TABLE 14.1-4.1: SUMMARY OF SUBJECT SURGICAL FEAR QUESTIONNAIRE – EFFICACY ANALYSIS SET | 50 |
| TABLE 14.1-4.2: SUMMARY OF SUBJECT SURGICAL FEAR QUESTIONNAIRE – SENSITIVITY ANALYSIS SET | 51 |
| TABLE 14.1-4.3: SUMMARY OF SUBJECT SURGICAL FEAR QUESTIONNAIRE – SAFETY ANALYSIS SET | 51 |
| TABLE 14.1-5.1: SUMMARY OF SURGERY CHARACTERISTICS – EFFICACY ANALYSIS SET | 52 |
| TABLE 14.1-5.2: SUMMARY OF SURGERY CHARACTERISTICS – SENSITIVITY ANALYSIS SET | Г53 |
| TABLE 14.1-5.3: SUMMARY OF SURGERY CHARACTERISTICS – SAFETY ANALYSIS SET | 53 |
| TABLE 14.1-6.1: INCIDENCE OF INTRAOPERATIVE MEDICATIONS - EFFICACY ANALYSIS SET | 54 |
| TABLE 14.1-6.2: INCIDENCE OF INTRAOPERATIVE MEDICATIONS - SAFETY ANALYSIS SET | 54 |
| TABLE 14.2-1.1A: ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 55 |
| TABLE 14.2-1.1B: SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72-EFFICACY ANALYSIS SET | 56 |
| TABLE 14.2-1.2A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY AGE – EFFICACY ANALYSIS SET | 57 |
| TABLE 14.2-1.2B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY AGE – EFFICACY ANALYSIS SET | 58 |
| TABLE 14.2-1.3A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY RACE – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.3B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY RACE – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.4A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY BMI STATUS – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.4B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY BMI STATUS – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.5A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY NUMBER OF PRIOR C-SECTIONS – EFFICACY ANALYSIS SET | 59 |

| TABLE 14.2-1.5B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY NUMBER OF PRIOR C-SECTIONS – EFFICACY ANALYSIS SET | 59 |
|---|---|
| TABLE 14.2-1.6A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY DISCHARGE TIME – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.6B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY DISCHARGE TIME – EFFICACY ANALYSIS SET | 59 |
| TABLE 14.2-1.7A: SUBGROUP ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY ANXIETY MEDICAL HISTORY – EFFICACY ANALYSIS SET | 60 |
| TABLE 14.2-1.7B: SUBGROUP SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS BY ANXIETY MEDICAL HISTORY – EFFICACY ANALYSIS SET | 60 |
| TABLE 14.2-1.8A: ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS – | 60 |
| TABLE 14.2-1.8B: SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 72 HOURS - | 60 |
| TABLE 14.2-2A: ANALYSIS OF AVERAGE ITCHING SCORES THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 61 |
| TABLE 14.2-2B: SUMMARY OF AVERAGE ITCHING SCORES THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 62 |
| TABLE 14.2-3.1A: ANALYSIS OF AVERAGE POSTSURGICAL ITCHING SCORES THROUGH 12, 24 AND 48 HOURS - EFFICACY ANALYSIS SET | 63 |
| TABLE 14.2-3.1B: SUMMARY OF AVERAGE POSTSURGICAL ITCHING SCORES THROUGH 12, 24 AND 48 HOURS - EFFICACY ANALYSIS SET | ,<br>64 |
| TABLE 14.2-3.2A: ANALYSIS OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 24<br>AND 48 HOURS, DAY 7 (168 HOURS) AND DAY 14 (336 HOURS) - EFFICACY<br>ANALYSIS SET | 65 |
| TABLE 14.2-3.2B: SUMMARY OF TOTAL OPIOID CONSUMPTION (OMED MG) THROUGH 24<br>AND 48 HOURS, DAY 7 (168 HOURS) AND DAY 14 (336 HOURS) - EFFICACY<br>ANALYSIS SET | 66 |
| TABLE 14.2-3.3A1: ANALYSIS OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 72<br>HOURS AFTER SURGERY OR HOSPITAL DISCHARGE WHICHEVER OCCURS<br>FIRST (GENERAL PAIN) - EFFICACY ANALYSIS SET | 67 |
| TABLE 14.2-3.3B1: SUMMARY OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 72<br>HOURS AFTER SURGERY OR HOSPITAL DISCHARGE WHICHEVER OCCURS<br>FIRST (GENERAL PAIN) – EFFICACY ANALYSIS SET | 68 |
| TABLE 14.2-3.4A1: ANALYSIS OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 24<br>AND 48 (GENERAL PAIN) - EFFICACY ANALYSIS SET | 69 |
| TABLE 14.2-3.4B1: SUMMARY OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 24<br>AND 48 (GENERAL PAIN) - EFFICACY ANALYSIS SET | 70 |
| TABLE 14.2-3.3A2: ANALYSIS OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 72<br>HOURS AFTER SURGERY OR HOSPITAL DISCHARGE WHICHEVER OCCURS<br>FIRST (PAIN AT INCISION SITE) - EFFICACY ANALYSIS SET | 71 |


| TABLE 14.2-3.3B2: SUMMARY OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 72 HOURS AFTER SURGERY OR HOSPITAL DISCHARGE WHICHEVER OCCURS FIRST (PAIN AT INCISION SITE) – EFFICACY ANALYSIS SET | 71 |
|---|---|
| TABLE 14.2-3.4A2: ANALYSIS OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 24 AND 48 (PAIN AT INCISION SITE) - EFFICACY ANALYSIS SET | 71 |
| TABLE 14.2-3.4B2: SUMMARY OF AVERAGE VAS PAIN INTENSITY SCORES THROUGH 24 AND 48 (PAIN AT INCISION SITE) - EFFICACY ANALYSIS SET | 71 |
| TABLE 14.2-3.5: ANALYSIS OF POSTSURGICAL OPIOID-FREE AND OPIOID-SPARING SUBJECTS THROUGH 72 HOURS - EFFICACY ANALYSIS SET | 72 |
| TABLE 14.2-3.6A: ANALYSIS OF OPIOID RELATED SYMPTOM DISTRESS SCALE (ORSDS) AT 12, 24, 48 AND 72 HOURS - EFFICACY ANALYSIS SET | 73 |
| TABLE 14.2-3.6B: SUMMARY OF OPIOID RELATED SYMPTOM DISTRESS SCALE (ORSDS) AT 12, 24, 48 AND 72 HOURS - EFFICACY ANALYSIS SET | 74 |
| TABLE 14.2-3.7A: ANALYSIS OF SUBJECTS MEETING MODIFIED POST ANESTHESIA DISCHARGE SCORING SYSTEM (MPADSS) CRITERIA FOR DISCHARGE READINESS AT 12, 24, 48 AND 72 HOURS - EFFICACY ANALYSIS SET | 75 |
| TABLE 14.2-3.7B: SUMMARY OF SUBJECTS MEETING MODIFIED POST ANESTHESIA DISCHARGE SCORING SYSTEM (MPADSS) CRITERIA FOR DISCHARGE READINESS AT EACH ASSESSED TIMEPOINT – EFFICACY ANALYSIS SET | 76 |
| TABLE 14.2-3.8: SUMMARY OF OVERALL ASSESSMENT OF SUBJECT'S SATISFACTION WITH PAIN CONTROL AT 72 HOURS OR HOSPITAL DISCHARGE, WHICHEVER OCCURS FIRST AFTER SURGERY – EFFICACY ANALYSIS SET | H<br>77 |
| TABLE 14.2-3.9: SUMMARY OF RECOVERY FROM CAESAREAN SECTION SCALE AT 24, 48, AND 72 HOURS OR HOSPITAL DISCHARGE, WHICHEVER COMES FIRST – EFFICACY ANALYSIS SET | 78 |
| TABLE 14.2-4.1A: ANALYSIS OF TOTAL POSTSURGICAL OPIOID CONSUMPTION (MG) IN MORPHINE EQUIVALENTS THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 81 |
| TABLE 14.2-4.1B: SUMMARY OF TOTAL POSTSURGICAL OPIOID CONSUMPTION (MG) IN MORPHINE EQUIVALENTS THROUGH 72 HOURS – EFFICACY ANALYSIS SET | 82 |
| TABLE 14.2-4.2: SUMMARY OF LENGTH OF HOSPITAL STAY – EFFICACY ANALYSIS SET | 83 |
| TABLE 14.2-4.3: SUMMARY OF NUMBER OF UNSCHEDULED PHONE CALLS OR OFFICE VISI<br>RELATED TO PAIN FROM DISCHARGE THROUGH DAY 14 – EFFICACY | |
| ANALYSIS SET | 84 |
| TABLE 14.2-4.4: SUMMARY OF NUMBER OF EMERGENCY DEPARTMENT (ED) VISITS – EFFICACY ANALYSIS SET | 85 |
| TABLE 14.2-4.5: ANALYSIS OF SUBJECTS WITH PERSISTENT OPIOID USE AT DAY 30 - EFFICACY ANALYSIS SET | 86 |
| TABLE 14.2-4.6A: ANALYSIS OF TIME SPENT IN POST-ANESTHESIA-CARE UNIT (PACU) – EFFICACY ANALYSIS SET | 87 |
| TABLE 14.2-4.6B: SUMMARY OF TIME SPENT IN POST-ANESTHESIA-CARE UNIT (PACU) – EFFICACY ANALYSIS SET | 88 |
| TABLE 14.2-4.7: ANALYSIS OF TIME TO FIRST UNASSISTED AMBULATION - EFFICACY ANALYSIS SET | 89 |
| TABLE 14.2-4.8: SUMMARY OF TIME TO FIRST BOWEL MOVEMENT - EFFICACY ANALYSIS SET | 90 |


402-C-414 (C-section TAP) Statistical Analysis Plan

| TABLE 14.3-1.1: OVERVIEW OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) - SAFETY ANALYSIS SET | 91 |
|---|---|
| TABLE 14.3-1.2.1: SUMMARY OF INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) BY PREFERRED TERM - SAFETY ANALYSIS SET | 92 |
| TABLE 14.3-1.2.2: SUMMARY OF SUBJECT INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) BY SYSTEM ORGAN CLASS AND PREFERRED TERM - SAFETY ANALYSIS SET | 93 |
| TABLE 14.3-1.3: SUMMARY OF SUBJECT INCIDENCE OF TREATMENT-EMERGENT ADVERSI<br>EVENTS (TEAES) BY SYSTEM ORGAN CLASS, PREFERRED TERM, AND WORST<br>SEVERITY - SAFETY ANALYSIS SET | |
| TABLE 14.3-1.4: SUMMARY OF SUBJECT INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS (TEAES) BY SYSTEM ORGAN CLASS, PREFERRED TERM, AND STRONGEST RELATIONSHIP TO STUDY DRUG - SAFETY ANALYSIS SET | E<br>95 |
| TABLE 14.3-1.5: SUMMARY OF SUBJECT INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS OF SPECIAL INTEREST (TEAESI) BY PREFERRED TERM - SAFETY ANALYSIS SET | E<br>96 |
| TABLE 14.3-2: SUMMARY OF VITAL SIGNS BY TIMEPOINT – SAFETY ANALYSIS SET | 97 |
| TABLE 14.3-3.1: INCIDENCE OF PRIOR MEDICATIONS – SAFETY ANALYSIS SET | 98 |
| TABLE 14.3-3.2: INCIDENCE OF CONCOMITANT MEDICATIONS – SAFETY ANALYSIS SET | 98 |


Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.1-1: Summary of Subject Disposition - All Screened Subjects

Site: Overall

| | 150 mcg | EXPAREL+50mcg | EXPAREL | _ |
|---|---|---|---|---|
| | Duramorph (SOC) | Duramorph | (N=XX) | Total |
| | (N=XX) | (N=XX) | n (응) | (N=XX) |
| | n (%) | n (응) | | n (%) |
| Screened [1] | | | | XX |
| Screen Failure | | | | xx (xx.x) |
| Enrolled | | | | xx (xx.x) |
| Randomized | XX | XX | xx | xx |
| Not Treated | xx | XX | XX | XX |
| Treated | XX | XX | XX | XX |
| TAP Infiltration Error per Ultrasound Image | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Safety Analysis Set [2]# | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Efficacy Analysis Set [3]@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol | | | | |
| Enrolled under Protocol Amendment2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Enrolled under Protocol Amendment1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Enrolled under Original Protocol | | | | |
| Completed Study@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from Study@ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons for Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of Efficacy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

402-C-414 (C-section TAP) Statistical Analysis Plan

**Note to programmer:** First page will present overall sites; subsequent pages will present each site - one site per page. For reasons for discontinuation only those reasons that appear in the data will appear on the table. For individual sites the label should be the site number. For the footnotes "Subjects treated with..." if no subjects were mistreated, then omit footnote.

<sup>[1]</sup> Signed the informed consent form [2] Received study drug [3] Received study drug and surgery Percentages for screen failure and enrolled based on number screened; others on number randomized.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Table 14.1-2.1: Summary of Subject Demographics - Efficacy Analysis Set

Site: Overall

| | Statistic | 150 mcg | EXPAREL+50mcg | EXPAREL | |
|---|---|---|---|---|---|
| | | Duramorph (SOC) | Duramorph | (N=XX) | |
| | | (N=XX) | (N=XX) | n (%) | Total |
| | | n (%) | n (%) | | (N=XX) |
| ge (yrs) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | XX, XX |
| ex | | | | | |
| Female | n (응) | | | | |
| _ | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Male | n (응) | | | | |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| thnicity | | | | | |
| Hispanic or Latino | n (%) | | | | |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Not Hispanic or Latino | n (%) | | , | , | , |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| ace | | | | | |
| American Indian/Alaska Native | n (응) | | | | |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Black/African American | n (%) | , | , | , | , |
| | (0.) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Asian | n (응) | | / | | |
| White | n /9-\ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| MUTTE | n (응) | ~~ (~~ ~) | · | · / · / · | .,,, /.,,, |
| Native Hawaiian/Pacific | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| · · · | 11 (6) | ( | / | () | / |
| slander | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |

Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

**Note to programmer:** Only categories available in the data will appear on the table. First page will present overall sites; subsequent pages will present each site - one site per page. For individual sites the label should be the site number.

Use this mock-up also for table:

Table 14.1-2.2: Summary of Subject Demographics - Sensitivity Analysis Set

Table 14.1-2.3: Summary of Subject Demographics - Safety Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.1-3.1: Summary of Subject Baseline Characteristics - Efficacy Analysis Set

| able 14.1-3.1: Summary of Subject Baseline Characteristics - Efficacy Analysis Set | | | | | |
|---|---|---|---|---|---|
| | | 150 mcg | EXPAREL+50mcg | | |
| | | Duramorph (SOC) | Duramorph | EXPAREL | Total |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XXX) |
| ASA Class | 2 - n (%) | XX | XX | XX | XX |
| | 3 − n (%) | XX.X | XX.X | XX.X | xx.x |
| | 4 - n (%) | X.XX | X.XX | X.XX | X.XX |
| | | XX.X | xx.x | XX.X | XX.X |
| | | XX, XX | XX, XX | XX, XX | xx, xx |
| ICG | | | | | |
| Interpretation | Normal - n (%) | XX | XX | XX | XX |
| | Abnormal, NCS - n (%) | XX.X | XX.X | XX.X | XX.X |
| | Abnormal, CS - n (%) | X.XX | x.xx | X.XX | X.XX |
| | | XX.X | xx.x | XX.X | XX.X |
| | | xx, xx | XX, XX | xx, xx | XX, XX |
| Height (cm) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Weight (kg) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | x.xx | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| BMI (kg/m2) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX | XX, XX |

| | | 150 mcg | EXPAREL+50mcg | | |
|---|---|---|---|---|---|
| | | Duramorph (SOC) | Duramorph | EXPAREL | Total |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XXX) |
| )irect Bili | | XX | XX | | XX |
| (unit) | n | AA | 222 | xx | 2121 |
| (dili c) | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X . XX | x <b>.</b> xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | XX, XX |
| GT (unit) | n | XX | XX | 77 | XX |
| GI (UIIIC) | Mean | XX.X | XX.X | XX | XX.X |
| | Mean<br>SD | x.xx | X.XX | XX.X | x.xx |
| | Median | XX.X | XX.X | X.XX | xx.x |
| | | | | xx.x | |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| DH (unit) | n | xx | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| LT (unit) | n | XX | XX | XX | XX |
| | Mean | XX.X | xx.x | XX.X | XX.X |
| | SD | x.xx | x.xx | X.XX | X.XX |
| | Median | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | XX, XX |
| ST (unit) | n | XX | xx | XX | XX |
| | Mean | XX.X | xx.x | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX | x.xx |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | xx, xx | XX, XX |
| BUN (unit) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | <b>X.</b> XX | x.xx | x.xx | X.XX |

| | 150 mcg<br>Duramorph (SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX |

CS = clinically significant. NCS = not clinically significant.

Table 14.1-3.2: Summary of Subject Baseline Characteristics - Sensitivity Analysis Set

Table 14.1-3.3: Summary of Subject Baseline Characteristics - Safety Analysis Set

XX

of the operation

n

| | | 150 mcg | EXPAREL+50mcg | | |
|---|---|---|---|---|---|
| | | Duramorph (SOC) | Duramorph | EXPAREL | Total |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XXX) |
| 1. I am afraid of | | | | | |
| operation | n | XX | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | x.xx | x.xx | X.XX | X.XX |
| | Median | xx.x | xx.x | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| 2. I am afraid of the | | | | | |
| anesthesia | n | XX | XX | xx | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | x.xx | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx |
| 3. I am afraid of the pair | n | | | | |
| after the operation | n | xx | XX | XX | XX |
| 1111111111 | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | xx, xx | XX, XX |
| 4. I am afraid of the | | xx | xx | | XX |
| unpleasant side effects | | | | | |
| (like nausea) after the | | | | | |
| operation | n | | | XX | |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| 5. I am afraid my health will deteriorate because | | xx | xx | | xx |

| Pacira Pharmaceuticals, Inc. | 402-C-414 (C-section TAP) |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

| EXPAREL | | | | | atistical Analysis Plan |
|---|---|---|---|---|---|
| | Mean | xx.x | XX.X | XX.X | xx.x |
| | SD | X.XX | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| 6. I am afraid the | | XX | xx | | XX |
| operation will fail | n | | | XX | |
| | Mean | XX.X | xx.x | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | X.XX |
| | Median | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | xx, xx | XX, XX |
| 8. I am afraid of the long duration of the rehabilitation after the | 3 | xx | xx | | xx |
| operation | n | | | XX | |
| - | Mean | XX.X | xx.x | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX | XX, XX |

0 = not at all afraid, 10 = very afraid.

Table 14.1-4.2: Summary of Subject Surgical Fear Questionnaire - Sensitivity Analysis Set

Table 14.1-4.3: Summary of Subject Surgical Fear Questionnaire - Safety Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

| | | 150 mcg<br>Duramorph<br>(SOC) (N=XX) | EXPAREL+50mcg Duramorph (N=XX) | EXPAREL<br>(N=XX)<br>n (%) | Total |
|---|---|---|---|---|---|
| Characteristic | Statistic | n (%) | n (%) | 11 (%) | (N=XX) |
| Duration of Surgery (hours) | n | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Median | XX | XX | XX | XX |
| | Min, Max | xx, xx | XX, XX | xx, xx | xx, xx |
| Type of Anesthesia | | | | | |
| General | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Spinal | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | N (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Intraoperative Med Used | | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| CSE Anesthesia Performed | | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Epidural Component of CSE | | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note, epidural component question is a follow up when CSE answer is Yes.

402-C-414 (C-section TAP) Statistical Analysis Plan

## Use this mock-up also for tables:

Table 14.1-5.2: Summary of Surgery Characteristics - Sensitivity Analysis Set

Table 14.1-5.3: Summary of Surgery Characteristics - Safety Analysis Set

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-414 |
|---|---|---|
| Table 14.1-6.1: Incidence of | f Intraoperative Medications - Efficacy Analysis Set | |

| | 150 mcg | EXPAREL+50mcg | EXPAREL | |
|---|---|---|---|---|
| | Duramorph (SOC) | Duramorph | (N=XX) | Total |
| natomical Therapeutic Class (ATC) | (N=XX) | (N=XX) | n (%) | (N=XX) |
| Preferred Name | n (%) | n (%) | | n (%) |
| ubjects taking at least one | | | | |
| nedication | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN1.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| IC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN2.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PN2.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TC. | | | | |

Medications are coded using World Health Organization Drug Dictionary (WHODD September 2018).

Sorted by descending total incidence by ATC and preferred name within ATC.

Intraoperative medications are those indicated as such by the investigator.

Subjects using the same prior medication more than once are counted only once at each summary level.

Table 14.1-6.2: Incidence of Intraoperative Medications - Safety Analysis Set  ${\bf T}$ 

Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.2-1.1a: Analysis of Total Opioid Consumption (OMED mg) Through 72 hours - Efficacy Analysis Set

| | 150 mcg<br>Duramorph (SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| Statistic | n (%) | n (%) | 11 (%) |
| LS Mean [1] | xxx.x | xxx.x | xxx.x |
| Standard Error of LS Mean [1] | xxx.xx | xxx.xx | XXX.XX |
| % Reduction [2] | xxx.x | xxx.x | |
| LSM Treatment Difference [1][3] | | xx.x | XX.X |
| 95% Confidence Interval [1][3] P-value, 1-sided [1][3] | | (xx.x, xx.x)<br>0.xxx | (xx.x, xx.x)<br>0.xxx |

LS = Least Square; LSM2 = LS Means in SOC group; LSM1 = LS Means in Active group.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and site and covariates of age and height on total opioid consumption. Subjects without any opioid use are assigned a value of 0 mg for summaries.

<sup>[2] %</sup> Reduction in Total Opioid Dose is calculated as (LSM2-LSM1)/LSM2\*100%.

<sup>[3]</sup> Test of Ha: LSM (Active) < LSM (SOC).

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.2-1.1b: Summary of Total Opioid Consumption (OMED mg) Through 72- Efficacy Analysis Set

| | 150 mcg Duramorph | EXPAREL+50mcg | EXPAREL |
|-----------|-------------------|---------------|---------|
| | (SOC) | Duramorph | (N=XX) |
| | (N=XX) | (N=XX) | n (%) |
| Statistic | n (%) | n (%) | |
| n | XX | XX | XX |
| GeoMean | XX.X | XX.X | XX.X |
| CV% | x.xx | x.xx | x.xx |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

GeoMean = Geometric mean. CV% = Coefficient of variation (%).

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-1.2a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by Age - Efficacy Analysis Set

150 mcg EXPAREL+50mcg EXPAREL Duramorph (SOC) Duramorph (N=XX)(N=XX)(N=XX)n (응) Age Statistic n (%) n (%) <35 years LS Mean [1] XXX.X XXX.X XXX.X Standard Error of LS Mean [1] XXX.XX XXX.XX XXX.XX % Reduction [2] XXX.X XXX.X LSM Treatment Difference [1][3] XX.X XX.X 95% Confidence Interval [1][3] (xx.x, xx.x)(xx.x, xx.x)P-value, 1-sided [1][3] 0.xxx 0.xxx >= 35 years LS Mean [1] xxx.x xxx.x xxx.x Standard Error of LS Mean [1] XXX.XX XXX.XX XXX.XX % Reduction [2] xxx.x XXX.X LSM Treatment Difference [1][3] XX.X XX.X 95% Confidence Interval [1][3] (xx.x, xx.x)(xx.x, xx.x)P-value, 1-sided [1][3] 0.xxx 0.xxx

LS = Least Square; LSM2 = LS Means in SOC group; LSM1 = LS Means in Active group.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and covariates of age and height on total opioid consumption. Subjects without any opioid use are assigned a value of 0 mg for summaries.

<sup>[2] %</sup> Reduction in Total Opioid Dose is calculated as (LSM2-LSM1)/LSM2\*100%.

<sup>[3]</sup> Test Ha: LSM (Active) < LSM (SOC).

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Protocol: 402-C-414

Table 14.2-1.2b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 hours by Age - Efficacy Analysis Set

| | | 150 mcg Duramorph | EXPAREL+50mcg | EXPAREL |
|-------------|-----------|-------------------|---------------|---------|
| | | (SOC) | Duramorph | (N=XX) |
| | | (N=XX) | (N=XX) | n (%) |
| Age | Statistic | n (%) | n (%) | |
| <35 years | N | xx | XX | xx |
| | GeoMean | xxx.x | XXX.X | xxx.x |
| | CV% | xxx.xx | XXX.XX | XXX.XX |
| | Median | xxx.x | XXX.X | xxx.x |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| >= 35 years | N | xx | XX | XX |
| | GeoMean | xxx.x | XXX.X | xxx.x |
| | CV% | XXX.XX | XXX.XX | xxx.xx |
| | Median | XXX.X | XXX.X | xxx.x |
| | Min, Max | XX, XX | XX, XX | xx, xx |

GeoMean = Geometric mean. CV% = Coefficient of variation (%).

Use Table 14.2-1.3a and 1.3b shell for (see SAP Section 9.7.2.1.2 for subgroup categories)

Table 14.2-1.3a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by Race - Efficacy Analysis Set

Table 14.2-1.3b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 hours by Race - Efficacy Analysis Set

Table 14.2-1.4a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by BMI Status - Efficacy Analysis Set

Table 14.2-1.4b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 hours by BMI Status - Efficacy Analysis Set

Table 14.2-1.5a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by Number of Prior C-Sections - Efficacy Analysis Set

Table 14.2-1.5b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 hours by Number of Prior C-Sections - Efficacy Analysis Set

Table 14.2-1.6a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by Discharge Time - Efficacy Analysis Set

Table 14.2-1.6b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 hours by Discharge Time - Efficacy Analysis Set

402-C-414 (C-section TAP) Statistical Analysis Plan

Table 14.2-1.7a: Subgroup Analysis of Total Opioid Consumption (OMED mg) Through 72 hours by Anxiety Medical History - Efficacy Analysis Set

Table 14.2-1.7b: Subgroup Summary of Total Opioid Consumption (OMED mg) Through 72 Hours by Anxiety Medical History - Efficacy Analysis Set

Table 14.2-1.8a: Analysis of Total Opioid Consumption (OMED mg) Through 72 hours - Sensitivity Analysis Set

Table 14.2-1.8b: Summary of Total Opioid Consumption (OMED mg) Through 72 Hours - Sensitivity Analysis Set

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.2-2a: Analysis of Average Itching Scores Through 72 hours - Efficacy Analysis Set

| | 150 mcg<br>Duramorph (SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| Statistic | n (%) | n (응) | |
| LS Mean [1] | xxx.x | xxx.x | xxx.x |
| Standard Error of LS Mean [1] | XXX.XX | XXX.XX | XXX.XX |
| LSM Treatment Difference [1][2] | | xx.x | XX.X |
| 95% Confidence Interval [1][2] | | (xx.x, xx.x) | (xx.x, xx.x) |
| P-value, 1-sided [1][2] | | 0.xxx | 0.xxx |

<sup>[1]</sup> From the Mixed Models.

<sup>[2]</sup> Test of Ha: LSM (Active) < LSM (150 mcg Duramorph (SOC)).

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.2-2b: Summary of Average Itching Scores Through 72 hours - Efficacy Analysis Set

| | 150 mcg Duramorph | EXPAREL+50mcg | EXPAREL |
|-----------|-------------------|---------------|---------|
| | (SOC) | Duramorph | (N=XX) |
| | (N=XX) | (N=XX) | n (%) |
| Statistic | n (%) | n (%) | |
| n | xx | XX | XX |
| Mean | XX.X | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx |
| Median | xx | xx | xx |
| Min, Max | XX, XX | XX, XX | xx, xx |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.1a: Analysis of Average Postsurgical Itching Scores Through 12, 24 and 48 Hours - Efficacy Analysis Set

| Timepoint | Statistic | 150 mcg<br>Duramorph (SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| 12 hours | LS Mean [1] Standard Error of LS Mean LSM Treatment Difference [1] 95% Confidence Interval P-value, 1-sided [2] | xxx.x<br>xxx.xx | xxx.x<br>xxx.xx<br>xx.x<br>(xx.x, xx.x) | xxx.x<br>xxx.xx<br>xx.x<br>(xx.x, xx.x)<br>0.xxxx |

24 hours

48 hours

<sup>[1]</sup> From the MMRM with age, height, treatment, site, timepoint and treatment-by-timepoint as factors and subjects as repeated measure unit over timepoints.

<sup>[2]</sup> Test of Ha: LSM (Active) < LSM (150 mcg Duramorph [SOC]).

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.1b: Summary of Average Postsurgical Itching Scores Through 12, 24 and 48 hours - Efficacy Analysis Set

| | | 150 mcg<br>Duramorph (SOC) | EXPAREL+50mcg<br>Duramorph | EXPAREL (N=XX) |
|---|---|---|---|---|
| | | (N=XX) | (N=XX) | n (%) |
| Timepoint | Statistic | n (%) | n (%) | |
| 12 hours | n | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | xx.xx | xx.xx | XX.XX |
| | Median | XX | XX | XX |
| | Min, Max | XX, XX | xx, xx | xx, xx |

48 hours

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-411 Table 14.2-3.2a: Analysis of Total Opioid Consumption (OMED mg) Through 24 and 48 hours, Day 7 (168 hours) and Day 14 (336 hours) - Efficacy Analysis Set

| | Statistic | 150 mcg<br>Duramorph (SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| 24 hrs | LS Mean [1] | XXX.X | xxx.x | xxx.x |
| | Standard Error of LS Mean [1] | xxx.xx | XXX.XX | XXX.XX |
| | % Reduction [2] | | XXX.XX | XXX.XX |
| | LSM Treatment Difference [1][3] | | XX.X | XX.X |
| | 95% Confidence Interval [1][3] | | (xx.x, xx.x) | (xx.x, xx.x) |
| | P-value, 1-sided [1][3] | | 0.xxx | 0.xxx |
| 48 hrs | LS Mean [1] | XXX.X | XXX.X | xxx.x |
| | Standard Error of LS Mean [1] | xxx.xx | XXX.XX | XXX.XX |
| | % Reduction [2] | | XXX.XX | XXX.XX |
| | LSM Treatment Difference [1][3] | | XX.X | XX.X |
| | 95% Confidence Interval [1][3] | | (xx.x, xx.x) | (xx.x, xx.x) |
| | P-value, 1-sided [1][3] | | 0.xxx | 0.xxx |

. . .

Note to programmer: Time periods to appear on this table, in order, are 0-24 hrs, 0-48 hrs, Day 7 (168 hours) and Day 14 (336 hours). Do not split a time period statistics across pages.

LS = Least Square; LSM2 = LS Means in IR Bupivacaine group; LSM1 = LS Means in EXPAREL 266 mg group.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and site and covariates of age and height on total opioid consumption. Subjects without any opioid use are assigned a value of 0 mg for summaries.

<sup>[2] %</sup> Reduction in Total Opioid Dose is calculated as (LSM2-LSM1)/LSM2\*100%.

<sup>[3]</sup> Test of Ha: LSM (EXPAREL 266 mg) < LSM (IR Bupivacaine).

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-411 Table 14.2-3.2b: Summary of Total Opioid Consumption (OMED mg) Through 24 and 48 hours, Day 7 (168 hours) and Day 14 (336 hours) - Efficacy Analysis Set

| | | | EXPAREL+50mcg | EXPAREL |
|---------------|-----------|-------------------|---------------|---------|
| | | 150 mcg Duramorph | Duramorph | (N=XX) |
| | | (SOC) (N=XX) | (N=XX) | n (%) |
| Time Interval | Statistic | n (%) | n (%) | |
| 24 hrs | n | XX | XX | XX |
| | GeoMean | XXX.X | XXX.X | XXX.X |
| | CV% | XXX.XX | XXX.XX | XXX.XX |
| | Median | XXX.X | XXX.X | xxx.x |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| 48 hrs | n | xx | XX | XX |
| | GeoMean | XXX.X | xxx.x | xxx.x |
| | CV% | xxx.xx | xxx.xx | xxx.xx |
| | Median | xxx.x | XXX.X | xxx.x |
| | Min, Max | XX, XX | xx, xx | xx, xx |

. . .

GeoMean = Geometric mean. CV% = Coefficient of variation (%).

**Note to programmer:** Time periods to appear on this table, in order, are 0-24 hrs, 0-48 hrs, Day 7 (168 hours) and Day 14 (336 hours). Do not split a time period statistics across pages.

Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.3al: Analysis of Average VAS Pain Intensity Scores Through 72 Hours After Surgery or Hospital Discharge Whichever Occurs First (General Pain) - Efficacy Analysis Set

| Statistic | 150 mcg<br>Duramorph (SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mc<br>g Duramorph<br>(N=XX)<br>n (%) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| LS Mean [1] | XXX.X | XXX.X | XXX.X |
| Standard Error of LS Mean | xxx.xx | XXX.XX | XXX.XX |
| LSM Treatment Difference [1] | | XX.X | XX.X |
| 95% Confidence Interval [2] | | (xx.x, xx.x) | (xx.x, xx.x) |
| Noninferiority Test P-value, 1-sided | | 0.xxx | 0.xxx |
| Superiority Test P-value, 1-sided | | | |

LS = Least Squares;

Programming note: if Superiority test fails, ie, p>0.05, then keep non-inferiority test and remove superiority test. Otherwise, remove non-inferiority test and keep superiority test.

VAS = 10 cm visual analog scale for pain, where 0 = no pain and 10 = worst possible pain.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and site and covariates of age and height.

<sup>[2]</sup> The non-inferiority of Active to 150 mcg Duramorph (SOC) is demonstrated if the upper limit is  $\leq 0.5$ . The superiority is demonstrated if the upper limit is  $\leq 0.5$ .

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.3bl: Summary of Average VAS Pain Intensity Scores Through 72 Hours After Surgery or Hospital Discharge Whichever Occurs First (General Pain) - Efficacy Analysis Set

| | 150 mcg Duramorph<br>(SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| Statistic | n (%) | n (%) | |
| n | xx | xx | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | xx.xx | xx.xx |
| Median | xx | XX | XX |
| Min, Max | XX, XX | XX, XX | XX, XX |

Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.4al: Analysis of Average VAS Pain Intensity Scores Through 24 And 48 (General Pain) - Efficacy Analysis Set - Multiple Imputation Results

| Timepoint | Statistic | 150 mcg Duramorph<br>(SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| 24 hours | LS Mean [1] | xxx.x | xxx.x | xxx.x |
| | Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| | LSM Treatment Difference [1] | XX.X | XX.X | |
| | 95% Confidence Interval [2] | (xx.x, xx.x) | (xx.x, xx.x) | |
| | Noninferiority Test P-value, 1-sided | 0.xxx | 0.xxx | |
| | Superiority Test P-value, 1-sided | 0.xxx | 0.xxx | |
| 48 hours | LS Mean [1] | xxx.x | xxx.x | xxx.x |
| | Standard Error of LS Mean | xxx.xx | XXX.XX | XXX.XX |
| | LSM Treatment Difference [1] | | XX.X | XX.X |
| | 95% Confidence Interval [2] | | (xx.x, xx.x) | (xx.x, xx.x) |
| | Noninferiority Test P-value, 1-sided | | 0.xxx | 0.xxx |
| | Superiority Test P-value, 1-sided | | 0.xxx | 0.xxx |

LS = Least Squares;

Programming note: if Superiority test fails, ie, p>0.05, then keep non-inferiority test and remove superiority test. Otherwise, remove non-inferiority test and keep superiority test.

VAS = 10 cm visual analog scale for pain, where 0 = no pain and 10 = worst possible pain.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and site and covariates of age and height.

<sup>[2]</sup> The non-inferiority of Active to 150 mcg Duramorph (SOC) is demonstrated if the upper limit is  $\leq 0.5$ . The superiority is demonstrated if the upper limit is  $\leq 0.5$ .

Pacira Pharmaceuticals, Inc.

402-C-414 (C-section TAP)

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.4bl: Summary of Average VAS Pain Intensity Scores Through 24 and 48 (General Pain) - Efficacy Analysis Set

| | | 150 mcg | EXPAREL+50mcg | EXPAREL |
|------------------|-----------|-----------------|---------------|---------|
| | | Duramorph (SOC) | Duramorph | (N=XX) |
| | | (N=XX) | (N=XX) | n (응) |
| Timepoint | Statistic | n (%) | n (%) | |
| 2 <b>4</b> hours | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX | XX | XX |
| | Min, Max | XX, XX | xx, xx | XX, XX |

48 hours

402-C-414 (C-section TAP) Statistical Analysis Plan

Table 14.2-3.3a2: Analysis of Average VAS Pain Intensity Scores Through 72 Hours After Surgery or Hospital Discharge Whichever Occurs First (Pain at Incision Site) - Efficacy Analysis Set

Table 14.2-3.3b2: Summary of Average VAS Pain Intensity Scores Through 72 Hours After Surgery or Hospital Discharge Whichever Occurs First (Pain at Incision Site) - Efficacy Analysis Set

Table 14.2-3.4a2: Analysis of Average VAS Pain Intensity Scores Through 24 And 48 (Pain at Incision Site) - Efficacy Analysis Set - Multiple Imputation Results

Table 14.2-3.4b2: Summary of Average VAS Pain Intensity Scores Through 24 and 48 (Pain at Incision Site) - Efficacy Analysis Set

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-411 Table 14.2-3.5: Analysis of Postsurgical Opioid-Free and Opioid-Sparing Subjects Through 72 hours - Efficacy Analysis Set

| | Statistic | 150 mcg Duramorph (SOC) (N=XX) n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| pioid-free | | | | |
| No Opioid-Free Percentage [1] | (%) | XX.X | XX.X | XX.X |
| Opioid-Free Percentage | (%) | XX.X | XX.X | XX.X |
| | Odds Ratio [2] | XX.X | XX.X | |
| | 95% CI for Odds Ratio | (xx.x, xx.x) | (xx.x, xx.x) | |
| | P-value, 1-sided [3] | 0.xxxx | 0.xxxx | |
| pioid-sparing | | | | |
| No Opioid-sparing Percentage [1] | (%) | XX.X | XX.X | XX.X |
| Opioid-s <b>paring</b> Percentage | (%) | XX.X | XX.X | XX.X |
| | Odds Ratio [2] | | XX.X | xx.x |
| | 95% CI for Odds Ratio | | (xx.x, xx.x) | (xx.x, xx.: |
| | P-value, 1-sided [3] | | 0.xxxx | 0.xxxx |
| | P-value, 1-sided [3] | | 0.xxxx | 0.xxxx |

<sup>[1]</sup> LS Means probability from the logistic regression with treatment, site, age, and height as explanatory variables.

<sup>[2]</sup> OR of Active over SOC.

<sup>[3]</sup> Test of Ha: Odds Ratio >1.
402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Protocol: 402-C-414

Table 14.2-3.6a: Analysis of Opioid Related Symptom Distress Scale (ORSDS) at 12, 24, 48 and 72 hours - Efficacy Analysis Set

Composite Score

| | | 150 mcg<br>Duramorph (SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| Timepoint | Statistic | n (응) | n (%) | |
| 12 hours | LS Mean [1] | xxx.x | xxx.x | xxx.x |
| | Standard Error of LS Mean LSM Treatment Difference [1] | XXX.XX | xxx.xx<br>xx.x | xxx.xx<br>xx.x |
| | 95% Confidence Interval P-value, 1-sided [2] | | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx |

24 hours

48 hours

72 hours

Note to programmer: Timepoints to appear on this table, in order, are 24, 48 and 72 hours.

First page is Composite Score, followed by Fatigue Score, Drowsiness Score, Inability to Concentration Score, Nausea Score, Constipation Score, Itching ..., Difficult with Urination Score, Confusion Score, and Retching/Vomiting Score.

Each symptom score is the average of frequency, severity, and botherness dimension scores.

Do not split a question's statistics across pages.

<sup>[1]</sup> From a Mixed Models with main effects of treatment visit and treatment by visit as covariates.

<sup>[2]</sup> Test of Ha: LSM (Active) < LSM (SOC). For Question 7 score, Test of Ha: LSM (Active) > LSM (SOC).

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Protocol: 402-C-414

Table 14.2-3.6b: Summary of Opioid Related Symptom Distress Scale (ORSDS) at 12, 24, 48 and 72 hours - Efficacy Analysis Set

## Composite Score

| Timepoint | Statistic | 150 mcg<br>Duramorph (SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| 24 hours | n<br>Mean | xx<br>xx.x | xx<br>xx.x | xx<br>xx.x |
| | SD<br>Median | xx.xx<br>xx | xx.xx<br>xx | XX.XX<br>XX |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| 18 hours | | | | |
| 7 <b>2</b> hours | | | | |

Repeat for symptom scores

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.7a: Analysis of Subjects Meeting Modified Post Anesthesia Discharge Scoring System (MPADSS) Criteria for Discharge Readiness at 12, 24, 48 and 72 hours - Efficacy Analysis Set

| Time Point | | 150 mcg<br>Duramorph (SOC) | EXPAREL+50mcg Duramorph | EXPAREL (N=XX) |
|---|---|---|---|---|
| | | (N=XX) | (N=XX) | n (%) |
| - | Statistic | n (응) | n (%) | |
| 24 | Odds Ratio [3]<br>95% CI for Odds Ratio<br>P-value, 1-sided [4] | xx.xx<br>xx.xxx<br>0.xxxx | xx.xx<br>xx.xxx | |
| Etc. | Odds Ratio<br>95% CI for Odds Ratio<br>P-value, 1-sided | | xx.xx<br>xx.xx<br>0.xxxx | xx.xx<br>xx.xxx<br>0.xxxx |

Note to programmer: Repeat for all valid Time periods for which data is available. Do not split a time period statistics across pages.

<sup>[1]</sup> Discharge-ready criterion is the MPADSS total score ≥9. Subjects who did not have assessment are considered "not ready".

<sup>[2]</sup> LS Means probability from the logistic regression with treatment, site, age, and height as explanatory variables.

<sup>[3]</sup> Ratio of Active over SOC in the odds of having 0 phone call.

<sup>[4]</sup> Test of Ha: Odds Ratio >1

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.7b: Summary of Subjects Meeting Modified Post Anesthesia Discharge Scoring System (MPADSS) Criteria for Discharge Readiness at Each Assessed Timepoint - Efficacy Analysis Set

| Time Point | | 150 mcg Duramorph<br>(SOC)<br>(N=XX) | EXPAREL+50mcg<br>Duramorph<br>(N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| | Statistic | n (%) | n (%) | 11 (0) |
| 24 | Criterion Met [1] (%) Criterion not Met (%) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Etc. | Criterion Met (%) Criterion not Met (%) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

<sup>[1]</sup> Discharge-ready criterion is the MPADSS total score ≥9. Subjects who did not have assessment are considered "not ready".

Note to programmer: Repeat for all valid Time periods for which data is available. Do not split a time period statistics across pages.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-3.8: Summary of Overall Assessment of Subject's Satisfaction with Pain Control at 72 hours or Hospital Discharge, Whichever Occurs First After Surgery - Efficacy Analysis Set

| | | 150 mcg<br>Duramorph | EXPAREL+50mcg<br>Duramorph | EXPAREL (N=XX) |
|---|---|---|---|---|
| | | (SOC) (N=XX) | (N=XX) | n (%) |
| Score | Statistic | n (%) | n (%) | |
| Summary | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | P-value, 2-sided[1] | 0.xxxx | 0.xxxx | |
| Score | | | | |
| 1: Extremely dissatisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2: Dissatisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3: Neither satisfied nor dissatisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4: Satisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5: Extremely Satisfied | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> P-value from CMH test performed using the "scores=modridit" option with site as stratification

**Note to programmer:** include all subjects at 72 hours after surgery (or at hospital discharge if earlier than 72 hours).

Table 14.2-3.9: Summary of Recovery from Caesarean Section Scale at 24, 48, and 72 Hours or Hospital Discharge, Whichever Comes First - Efficacy Analysis Set

| | | 150 mcg<br>Duramorph | EXPAREL+50mcg Duramorph | EXPAREL (N=XX) |
|---|---|---|---|---|
| Question | Statistic | (SOC) (N=XX)<br>n (%) | (N=XX)<br>n (%) | n (%) |
| Question | Statistic | 11 (10) | 11 (**) | |
| 1. I recovered quickly from my cesarean | n | XX | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX |
| 2. I was able to get out of bed soon | | | | |
| after my cesarean | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| 3. My mobility was seriously affected | | XX | XX | |
| by the cesarean | n | | | XX |
| | Mean | xx.x | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| 4. The cesarean interfered with my | | xx | xx | |
| ability to care for my baby | n | | | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | x.xx |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| 5. The cesarean prevented me from | n | xx | xx | XX |

| | | 150 mcg | EXPAREL+50mcg | EXPAREL |
|---|---|---|---|---|
| | | Duramorph | Duramorph | (N=XX) |
| Question | Statistic | (SOC) $(N=XX)$ | (N=XX) | n (%) |
| feeding my baby | Statistic | n (%) | n (%) | |
| reeding my baby | | XX.X | XX.X | |
| | Mean | | | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| 6. I was able to change my baby soon | | xx | xx | |
| after the cesarean | n | | | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | x.xx | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| 7. I was able to care for my own | | XX | XX | |
| nygiene needs soon after surgery | n | | | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| 3. The pain from the surgery prevented | | xx | xx | |
| me from doing what I wanted | n | | | XX |
| - | Mean | XX.X | XX.X | XX.X |
| | SD | x.xx | X.XX | x.xx |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| I was tired for a long time after | | XX | XX | |
| surgery | n | | | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |

402-C-414 (C-section TAP) Statistical Analysis Plan

| Question | Statistic | 150 mcg<br>Duramorph<br>(SOC) (N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | xx, xx |

<sup>0 =</sup> strongly disagree and 7 = strongly agree.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-4.1a: Analysis of Total Postsurgical Opioid Consumption (mg) in Morphine Equivalents Through 72 hours - Efficacy Analysis Set

| Statistic | 150 mcg<br>Duramorph (SOC)<br>(N=XX)<br>n (%) | EXPAREL+50mc<br>g Duramorph<br>(N=XX)<br>n (%) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| LS Mean [1] | xxx.x | xxx.x | xxx.x |
| Standard Error of LS Mean | XXX.XX | XXX.XX | XXX.XX |
| LSM Treatment Difference [1] | | XX.X | XX.X |
| 95% Confidence Interval [2] | | (xx.x, xx.x) | (xx.x, xx.x) |
| Noninferiority Test P-value, 1-sided Superiority Test P-value, 1-sided | | 0.xxx | 0.xxx |

LS = Least Square;

Programming note: if Superiority test fails, ie, p>0.05, then keep non-inferiority test and remove superiority test. Otherwise, remove non-inferiority test and keep superiority test.

<sup>[1]</sup> From an ANCOVA with main effects of treatment and site and covariates of age and height.

<sup>[2]</sup> The non-inferiority of Active to 150 mcg Duramorph (SOC) is demonstrated if the upper limit on logarithm scale is <=0.8. The superiority is demonstrated if the upper limit is <0.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-4.1b: Summary of Total Postsurgical Opioid Consumption (mg) in Morphine Equivalents Through 72 hours - Efficacy Analysis Set

| | 150 mcg Duramorph<br>(SOC)<br>(N=XX) | EXPAREL+50mcg Duramorph (N=XX) | EXPAREL<br>(N=XX)<br>n (%) |
|---|---|---|---|
| Statistic | n (%) | n (%) | |
| n | xx | xx | xx |
| GeoMean | xx.x | xx.x | xx.x |
| CV% | XX.XX | xx.xx | xx.xx |
| Median | xx | XX | XX |
| Min, Max | XX, XX | XX, XX | XX, XX |

GeoMean = Geometric mean. CV% = Coefficient of variation (%).

402-C-414 (C-section TAP) Pacira Pharmaceuticals, Inc. **EXPAREL** 

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-411 Table 14.2-4.2: Summary of Length of Hospital Stay - Efficacy Analysis Set 150 mcg Duramorph EXPAREL EXPAREL+ (SOC) 50mcg Duramorph (N=XX)(N=XX)(N=XX)n (%) Statistic n (%) n (%) Ν XX XX XX Mean XXX.X XXX.X XXX.X SD XXX.XX XXX.XX XXX.XX Median XXX.X XXX.X XXX.X Min, Max XX, XX XX, XX XX, XX

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-411

Table 14.2-4.3: Summary of Number of Unscheduled Phone Calls or Office Visits Related to Pain from Discharge Through Day 14 - Efficacy Analysis Set

| | 150 mcg Duramorph (SOC) | EXPAREL+50mcg Duramorph | EXPAREL |
|-----------|-------------------------|-------------------------|---------|
| | (N=XX) | (N=XX) | (N=XX) |
| Statistic | n (%) | n (%) | n (%) |
| N | xx | xx | XX |
| Mean | XXX.X | xxx.x | xxx.x |
| SD | xxx.xx | xxx.xx | xxx.xx |
| Median | XXX.X | xxx.x | xxx.x |
| Min, Max | XX, XX | XX, XX | xx, xx |

402-C-414 (C-section TAP) Statistical Analysis Plan

| (ED) Visits - Efficacy Analys<br>+50mcg Duramorph<br>(N=XX)<br>n (%) | sis Set EXPAREL (N=XX) n (%) |
|---|---|
| (N=XX) | (N=XX) |
| , | , |
| n (%) | n (%) |
| XX | XX |
| XXX.X | XXX.X |
| XXX.XX | xxx.xx |
| VVV V | XXX.X |
| AAA • A | XX, XX |
| | xxx.x |

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmaceuticals | | (Page X of Y) | Protocol: | 402-C-414 |
|---|---|---|---|---|
| Table 14.2-4.5: Analysis o | f Subjects with Persi | stent Opioid Use at Day 30 - Effi | icacy Analysis Set | |
| | 150 mcg Duramorph | EXPAREL+50mcg Duramorph | EXPAREL | |
| | (SOC) (N=XX) | (N=XX) | (N=XX) | |
| | n (%) | n (%) | n (%) | |
| NO | XX.X | xx.x | xx.x | |
| Yes | xx.x | xx.x | xx.x | |

Note, persistent opioid use is defined for subjects who answered Yes to the question of opioid use at Day 30.

| Pacira Pharmaceuticals | (Page X of Y) | | Protocol: 402-C-411 |
|---|---|---|---|
| Table 14.2-4.6a: Analysis of Time Spent | in Post-Anesthesia-Care Uni | t (PACU) - Efficacy | y Analysis Set |
| | | EXPAREL+50mcg | EXPAREL |
| | 150 mcg Duramorph | Duramorph | (N=XX) |
| | (SOC) (N=XX) | (N=XX) | n (%) |
| Statistic | n (%) | n (응) | |
| LS Mean [1] | XXX.X | 777 V | VVV V |
| 2 3 | | XXX.X | XXX.X |
| Standard Error of LS Mean [1] | XXX.XX | XXX.XX | XXX.XX |
| LSM Treatment Difference [1][2] | | XX.X | XX.X |
| 95% Confidence Interval [1][2] | | (xx.x, xx.x) | (xx.x, xx.x) |
| P-value, 1-sided [1][2] | | 0.xxxx | 0.xxxx |

<sup>[1]</sup> From the gamma (or normal) distribution and log link function and main effects of treatment and site and covariates of age and height on time spent in PACU.

<sup>[2]</sup> Test of Ha: LSM (Active) < LSM (150 mcg Duramorph (SOC)).

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmace | euticals | (Page X of Y) | Protocol: 402-C-411 |
|---|---|---|---|
| Table 14.2-4.6k | o: Summary of Time Spent in Post | t-Anesthesia-Care Unit (PACU) - E | Efficacy Analysis Set |
| | 150 mcg Duramorph (SOC) | EXPAREL+50mcg Duramorph | EXPAREL |
| | (N=XX) | (N=XX) | (N=XX) |
| Statistic | n (%) | n (%) | n (%) |
| N | xx | xx | xx |
| Mean | xxx.x | xxx.x | XXX.X |
| SD | XXX.XX | XXX.XX | xxx.xx |
| Median | XXX.X | XXX.X | XXX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.2-4.7: Analysis of Time to First Unassisted Ambulation - Efficacy Analysis Set

| | Statistic | 150 mcg Duramorph (SOC) (N=XX) n (%) | EXPAREL+50mcg<br>Duramorph (N=XX)<br>n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| -72 hours | | | | |
| Number of Subjects with | | | | |
| Ambulation (observed) | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No Ambulation (censored) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to Ambulation | | | | |
| Quartiles [1] | | | | |
| First (25% Ambulated) | Estimate | xx.xx | xx.xx | XX.XX |
| | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Median (50% Ambulated) | Estimate | xx.xx | xx.xx | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75% Ambulated) | Estimate | xx.xx | XX.XX | xx.xx |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | XX.XX | xx.xx | XX.XX |
| Maximum | Observed | xx.xx* | xx.xx* | xx.xx |
| Log-rank p-value, 2-sided | | | | |
| Cox regression Hazard Ratio[2] | Estimate | xx.xx | xx.xx | xx.xx |
| P-value, 2-sided | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx)<br>0.xxxx | (xx.xx, xx.xx)<br>0.xxxx |

<sup>\*</sup> indicates censored observation. CI = confidence interval

<sup>[1]</sup> Estimates from the Kaplan-Meier survival curve.

<sup>[2]</sup> P-value for the Active to SOC comparison using the Cox regression model with treatment and site as factors and age and height as covariates.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y)
Table 14.2-4.8: Summary of Time to First Bowel Movement - Efficacy Analysis Set

| | Statistic | 150 mcg Duramorph<br>(SOC) (N=XX)<br>n (%) | EXPAREL+50mcg<br>Duramorph (N=XX)<br>n (%) | EXPAREL (N=XX) n (%) |
|---|---|---|---|---|
| 0-72 hours | | | | |
| Number of Subjects with | | | | |
| Bowel Movement (observed) | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No Bowel Movement (censored) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to Bowel Movement | | | | |
| Quartiles [1] | | | | |
| First (25% Bowel Movement) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Median (50% Bowel Movement) | Estimate | XX.XX | XX.XX | XX.XX |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Third (75% Bowel Movement) | Estimate | XX.XX | XX.XX | xx.xx |
| | (95% CI) | (xx.xx,xx.xx) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Minimum | Observed | xx.xx | XX.XX | XX.XX |
| Maximum | Observed | xx.xx* | XX.XX* | xx.xx |
| Log-rank p-value, 2-sided | | | | |
| Cox regression Hazard Ratio[2] | Estimate | xx.xx | xx.xx | xx.xx |
| | (95% CI) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| P-value, 2-sided | • | | 0.xxxx | 0.xxxx |

<sup>\*</sup> indicates censored observation. CI = confidence interval

<sup>[1]</sup> Estimates from the Kaplan-Meier survival curve.

<sup>[2]</sup> P-value for the Active to SOC comparison using the Cox regression model with treatment and site as factors and age and height as covariates.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.3-1.1: Overview of Treatment-Emergent Adverse Events (TEAEs) - Safety Analysis Set

| | 150 mcg | EXPAREL+50mcg | EXPAREL | Total |
|---|---|---|---|---|
| | Duramorph (SOC) | Duramorph | (N=XX) | (N=XX) |
| | (N=XX) | (N=XX) | n (%) | n (%) |
| Number of | n (응) | n (%) | | |
| Subjects with Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Severity of Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At Least One Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At Least One Serious | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects Discontinued due to TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ied on Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to programmer: All categories on this table should appear, even if not present in the data.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.3-1.2.1: Summary of Incidence of Treatment-Emergent Adverse Events (TEAEs) by Preferred Term - Safety Analysis Set

| Preferred Term | 150 mcg<br>Duramorph<br>(SOC) (N=XX)<br>n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| Subjects with ≥1 TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 PT2 PT3 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA v21.1).

Sorted by descending order of Total incidence.

Subjects experiencing the same TEAE more than once are counted only once at each summary level.

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmaceuticals Table 14.3-1.2.2: Summary of Subject Incidence Class and Preferred Term - Safety Analysis Set | (Page X of Y)<br>e of Treatment-En | mergent Adverse Ev | | col: 402-C-414<br>y System Organ |
|---|---|---|---|---|
| | 150 mcg | EXPAREL+50mcg | EXPAREL | Total |
| | Duramorph | Duramorph | (N=XX) | (N=XX) |
| System Organ Class | (SOC) $(N=XX)$ | (N=XX) | n (%) | n (%) |
| Preferred Term | n (%) | n (%) | | |
| Subjects with ≥1 TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2.2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ETC. | , | , , | , , | , , |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA v21.1). Sorted by system organ class and preferred term in alphabetical order. Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.3-1.3: Summary of Subject Incidence of Treatment-Emergent Adverse Events (TEAEs) by System Organ

Class, Preferred Term, and Worst Severity - Safety Analysis Set

| System Organ Class<br>Preferred Term | Worst<br>Severity | 150 mcg Duramorph (SOC) (N=XX) n (%) | EXPAREL+50mcg Duramorph (N=XX) n (%) | EXPAREL (N=XX) n (%) | Total<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|
| Subjects with ≥1 TEAE | Mild | ( | ( | ( | ( |
| Subjects with it is | MIIG<br>Moderate | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.1 | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1.2 | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

. . .

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA v21.1). Sorted by descending order of Total incidence by system organ class and preferred term. Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Table 14.3-1.4: Summary of Subject Incidence of Treatment-Emergent Adverse Events (TEAEs) by System Organ Class, Preferred Term, and Strongest Relationship to Study Drug - Safety Analysis Set

| | | 150 mcg | EXPAREL+50mcg | EXPAREL | Total |
|---|---|---|---|---|---|
| | | Duramorph (SOC) | Duramorph | (N=XX) | (N=XX) |
| System Organ Class | Strongest | (N=XX) | (N=XX) | n (%) | n (%) |
| Preferred Term | Relation | n (응) | n (%) | | |
| Subjects with ≥1 TEAE | Not | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| | | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| SOC1 | Not | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| | | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| PT1.1 | Not | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| | | | | | XX |
| | Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA v21.1). Sorted by descending total incidence by system organ class and preferred term within system organ class. Subjects experiencing the same TEAE more than once are counted only once at each summary level. "Related" is "possible", "probable", or "definite" and "Not Related" is "unlikely" or "unrelated" by the investigator's assessment.

| Pacira Pharmaceuticals, Inc. | 402-C-414 (C-section TAP) |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

| Pacira Pharmaceuticals Table 14.3-1.5: Summary of Subject (TEAESI) by Preferred Term - Safety A | Incidence of Tr | X of Y)<br>reatment-Emergent | | Protocol: 402-C-414 Special Interest |
|---|---|---|---|---|
| | 150 mcg<br>Duramorph<br>(SOC) | EXPAREL+50mcg<br>Duramorph | EXPAREL<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| Group<br>Preferred Term | (N=XX)<br>n (%) | (N=XX)<br>n (%) | . , | . , |
| Subjects with ≥1 TEAESI | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| FALL | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cardiac TEAESI Angina Myocardial infarction | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Neurologic TEAESI Tinnitus Perioral numbness | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Adverse events coded using the Medical Dictionary for Regulatory Activities (MedDRA 21.1). Sorted by system organ class and preferred term in alphabetical order. Subjects experiencing the same TEAE more than once are counted only once at each summary level.

Note to programmer: see SAP the list of AESI

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Table 14.3-2: Summary of Vital Signs by Timepoint - Safety Analysis Set

| | 110020 | Rate (bpm) | 150 m<br>Duram<br>(SOC) | | EXPAREL+! Duramorp! (N=XX) | | EXPAREL (N=XX) n (%) | | Total |
|---|---|---|---|---|---|---|---|---|---|
| Timepoint | Value | Statistic | n (%) | (11 1111) | n (응) | | | | (N=XXX) |
| Baseline | Actual | n | | XX | | XX | | XX | XX |
| Dasciine | 7100001 | Mean | | XX.X | | XX.X | | XX.X | XX.X |
| | | SD | | X.XX | | x.xx | | X.XX | X.XX |
| | | Median | | XX.X | | XX.X | | XX.X | XX.X |
| | | Min, Max | XX, | | XX | , XX | XX, | XX | XX, XX |
| | Baseline | | | | | | | | |
| OR | [1] | n | | XX | | XX | | XX | XX |
| | | Mean | | xx.x | | XX.X | | xx.x | XX.X |
| | | SD | | x.xx | | X.XX | | X.XX | X.XX |
| | | Median | | XX.X | | XX.X | | XX.X | XX.X |
| | | Min, Max | XX, | XX | XX | , XX | XX, | XX | XX, XX |
| | Actual | n | | XX | | XX | | XX | XX |
| | | Mean | | XX.X | | XX.X | | XX.X | XX.X |
| | | SD | | x.xx | | X.XX | | x.xx | X.XX |
| | | Median | | XX.X | | XX.X | | XX.X | XX.X |
| | | Min, Max | XX, | XX | XX | , XX | XX, | XX | XX, XX |
| | Change | n | | XX | | XX | | XX | xx |
| | | Mean | | XX.X | | XX.X | | XX.X | XX.X |
| | | SD | | x.xx | | X.XX | | X.XX | X.XX |
| | | Median | | XX.X | | XX.X | | XX.X | XX.X |
| | | Min, Max | XX, | XX | XX | , XX | XX, | XX | xx, xx |

<sup>[1]</sup> Baseline (prior to surgery) for subjects with data at the timepoint.

402-C-414 (C-section TAP) Statistical Analysis Plan

Note to programmer: Vital signs are 'Resting Heart Rate (bpm)', 'Systolic Blood Pressure (mmHg)' and 'Diastolic Blood Pressure (mmHg)'. Timepoints to appear on this table are, in order of appearance, Baseline (prior to surgery), OR, PACU and Discharge. Do not split timepoint statistics across pages.

**Note to programmer:** Use mock-up 14.1-6.1 for tables:

Table 14.3-3.1: Incidence of Prior Medications - Safety Analysis Set.

On this table change the footnote 'Intraoperative medications are those indicated as such by the investigator' to read 'Prior medications are those stopped before start of study drug administration.'

Table 14.3-3.2: Incidence of Concomitant Medications - Safety Analysis Set.

On this table change the footnote 'Intraoperative medications are those indicated as such by the investigator' to read 'Concomitant medications are those taken after the start of study drug administration and are not designated intraoperative medications.'

## 17 LIST OF LISTINGS

| LISTING 16.2-1: SUBJECT DISPOSITION – ALL RANDOMIZED SUBJECTS | 101 |
|---|---|
| LISTING 16.2-2: RANDOMIZATION AND ANALYSIS SETS – ALL RANDOMIZED SUBJECTS | 102 |
| LISTING 16.2-3: INCLUSION/EXCLUSION CRITERIA – FAILURES – ALL RANDOMIZED SUBJECTS | 103 |
| LISTING 16.2-4: DEMOGRAPHICS – ALL RANDOMIZED SUBJECTS | 104 |
| LISTING 16.2-5: HEIGHT AND WEIGHT – ALL RANDOMIZED SUBJECTS | 105 |
| LISTING 16.2-6: SURGERY – ALL RANDOMIZED SUBJECTS | 106 |
| LISTING 16.2-7: VISUAL ANALOG SCALE (VAS) – ALL RANDOMIZED SUBJECTS | 107 |
| LISTING 16.2-8.1: POSTSURGICAL TOTAL OPIOID DOSE (OMED MG) AND OPIOID-FREE<br>STATUS – ALL RANDOMIZED SUBJECTS | 108 |
| LISTING 16.2-8.2: POSTSURGICAL OPIOID DOSING – ALL RANDOMIZED SUBJECTS | 109 |
| LISTING 16.2-9: PRESCRIPTION DAILY PAIN MEDICATION – ALL RANDOMIZED SUBJECTS | S110 |
| LISTING 16.2-10: RESCUE MEDIATION – ALL RANDOMIZED SUBJECTS | 111 |
| LISTING 16.2-11: OPIOID RELATED SYMPTOM DISTRESS SCALE (ORSDS) – ALL<br>RANDOMIZED SUBJECTS | 112 |
| LISTING 16.2-12.1: RECOVERY FROM CAESAREAN SECTION SCALE (RCSS) – QUESTION TEXT | 113 |
| LISTING 16.2-12.2: RECOVERY FROM CAESAREAN SECTION SCALE (RCSS) – ALL RANDOMIZED SUBJECTS | 114 |
| LISTING 16.2-13: MODIFIED POST-ANESTHESIA DISCHARGE SCORING SYSTEM (MPADSS<br>ALL RANDOMIZED SUBJECTS | ) –<br>115 |
| LISTING 16.2-14.1: SURGICAL FEAR QUESTIONNAIRE (SFQ) – QUESTION TEXT | 116 |
| LISTING 16.2-14.2: SURGICAL FEAR QUESTIONNAIRE (SFQ) – ALL RANDOMIZED SUBJECT | ΓS117 |
| LISTING 16.2-15: PULSE OXIMETRY (LOG FORM) – ALL RANDOMIZED SUBJECTS | 118 |
| LISTING 16.2-16: SUBJECT SATISFACTION WITH POST-SURGICAL PAIN CONTROL AT 72<br>HOURS – ALL RANDOMIZED SUBJECTS | 119 |
| LISTING 16.2-17: DAY 14 PHONE CALL – ALL RANDOMIZED SUBJECTS | 120 |
| LISTING 16.2-18: VITAL SIGNS ASSESSMENT – ALL RANDOMIZED SUBJECTS | 121 |
| LISTING 16.2-19: ELECTROCARDIOGRAM FINDINGS AT SCREENING – INVESTIGATOR<br>ASSESSMENT – ALL RANDOMIZED SUBJECTS | 122 |
| LISTING 16.2-20: PAIN INTENSITY SCALE- TIMEPOINT QUESTIONS – ALL RANDOMIZED SUBJECTS | 123 |
| LISTING 16.2-21: ASSESSMENT OF ITCHING – ALL RANDOMIZED SUBJECTS | 124 |
| LISTING 16.2-22.1: ALL ADVERSE EVENTS – ALL RANDOMIZED SUBJECTS | 125 |
| LISTING 16.2-22.2: TREATMENT-EMERGENT ADVERSE EVENTS – ALL RANDOMIZED SUBJECTS | 125 |
| LISTING 16.2-22.3: ALL SERIOUS ADVERSE EVENTS – ALL RANDOMIZED SUBJECTS | 125 |
| LISTING 16.2-22.4: TREATMENT-EMERGENT ADVERSE EVENTS OF SPECIAL INTEREST – ALL RANDOMIZED SUBJECTS | 125 |

| Pacira Pharmaceuticals, Inc. EXPAREL | 402-C-411 (C-section TAP)<br>Statistical Analysis Plan |
|---|---|
| LISTING 16.2-23.1: PRIOR MEDICATIONS – ALL RANDOMIZED SUBJECTS | 126 |
| LISTING 16.2-23.2: CONCOMITANT MEDICATIONS – ALL RANDOMIZED SUBJE | CTS 126 |
| LISTING 16.2-24: MEDICAL HISTORY/SURGERY – ALL SUBJECTS | 127 |
| LISTING 16.2-25: INTRAOPERATIVE MEDICATIONS – RANDOMIZED SUBJECTS | 128 |
| LISTING 16.2-26: STUDY DRUG ADMINISTRATION – RANDOMIZED SUBJECTS | 129 |
| LISTING 16.2-27: STANDARD OF CARE – RANDOMIZED SUBJECTS | 130 |
| LISTING 16.2-28: PHYSICAL EXAMINATION – RANDOMIZED SUBJECTS | 131 |
| LISTING 16.2-29: URINE DRUG SCREEN, ALCOHOL BLOOD TEST AND PREGNAL ALL SUBJECTS | NCY TEST – 132 |
| LISTING 16.2-30: ADMISSION AND DISCHARGE – RANDOMIZED SUBJECTS | 133 |
| LISTING 16.2-31: IMPORTANT PROTOCOL DEVIATIONS - RANDOMIZED SUBJE | CTS 134 |
| LISTING 16.2-32: ULTRASOUND COLLECTION – RANDOMIZED SUBJECTS | 135 |
| LISTING 16.2-33: UNIQUE ADVERSE EVENTS TERMS AND ASSOCIATED CODEI | D TERMS 136 |
| LISTING 16.2-34: UNIQUE MEDICATION TERMS AND ASSOCIATED CODED TERMS | RMS 137 |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-1: Subject Disposition - All Randomized Subjects

TREATMENT: treatment-name

Date of

Subject Last Visit (Day) End of Study Status Specify

XXX-YYYY DDMONYYYY (XX)

Note to programmer: End of study status for subject who early terminated from the study is the primary reason for termination. If subject discontinued due to an AE then the reason should read 'ADVERSE EVENT, AE # X'. If subject discontinued due to death the reason should read 'DEATH ON DDMONYYYY'. For those reasons that also collected a specify text, that text belongs in the specify column.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Listing 16.2-2: Randomization and Analysis Sets - All Randomized Subjects

| | Randomization | | | | |
|----------|-----------------|--------|------------|--------|----------|
| | | | Treatment | | |
| Subject | Date and Time | Number | Group | Safety | Efficacy |
| | | | EXPAREL+50 | | |
| | | | mcg | | |
| XXX-YYYY | DDMONYYYYTHH:MM | XXXXX | Duramorph | X | X |
| | | | EXPAREL | | |
| | | | SOC | | |

Note to programmer: Analysis set will by 'Y' if subject in set, blank otherwise.

402-C-414 (C-section TAP) Statistical Analysis Plan

| | | | • |
|---|---|---|---|
| | armaceuticals<br>6.2-3: Inclusion/E | | (Page X of Y)<br>on criteria - Failures - All Randomized Subjects |
| TREATMENT | : treatment-name | | |
| | | Protocol Versi | Lon |
| Subject | Visit | Enrolled Under | Criteria Not Met |
| XXX-YYYY | DDMONYYYY | Amendment 1 | xxxxxxxxx |
| | | Amendment 2 | |

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y)

Listing 16.2-4: Demographics - All Randomized Subjects

TREATMENT: treatment-name

| Subject | Initials | Birth Date | Age(yrs) | Sex | Race | Ethnicity | ASA Class |
|---|---|---|---|---|---|---|---|
| XXX-YYYY | AMZ | DDMONYYYY | XX | XXXXXX | XXXXXXXX | XXXXXXXX | X |

Note to programmer: If race is 'other' then race should be 'Other: other-specify-text'.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Listing 16.2-5: Height and Weight - All Randomized Subjects

Protocol: 402-C-414

TREATMENT: treatment-name

| Subject | Collection Date (Day) | Height (cm) | Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|
| XXX-YYYY | DDMONYYYYTHH:MM (-XX) | XXX.X | XXX.X | XX.X |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414
Listing 16.2-6: Surgery - All Randomized Subjects

TREATMENT: treatment-name

Intraoperat CSEPerforme Component ive d/ of CSE

| Subje<br>ct | Date<br>(Day) | Star<br>t<br>Time | Stop<br>Time | Durati<br>on<br>(hrs) | Locati<br>on | Incisi<br>on<br>Length<br>(cm) | SOC<br>Admi<br>n<br>Time | Anesthes<br>ia Type | Intraoperat<br>ive<br>Medications<br>Administere<br>d | CSEPerforme<br>d/ | Component<br>of CSE<br>Administer<br>ed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-<br>YYYY | DDMONYY<br>YY (XX) | НН:М<br>М | НН:М<br>М | Х.Х | XXXXX | XX.X | НН:М<br>М | | Yes | Yes | No |
| | | | | | | | | | No | Yes | Yes |

Note to programmer: If anesthesia type is 'other' then text should read 'other: specify-text'.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-7: Visual Analog Scale (VAS) - All Randomized Subjects

| TREATMENT: | treatment-name | | • | - | | |
|---|---|---|---|---|---|---|
| | | Time From Dos | e | | | |
| | | Scheduled | Actual | Deviation | VAS | Pain-Free |
| Subject | Date Time (Day) | (hr) | (hr) | (hrs) | (cm) | $(VAS \leq 1.5cm)$ |
| XXX-YYYY | DDMONYYYYTHH:MM (X) | XX.XX | XX.XX | XXXX | XX.X | Y |

VAS: 0=No pain to 10=Worst Pain Imaginable

ND=Not Done NA=Not Applicable

Protocol: 402-C-414

Note to programmer: Sort by VAS collection date and time. If VAS was taken due to rescue medication dosing, put RESCUE in scheduled column and hours from dose in actual column - leave deviation column blank. Do not split a subject's data across pages if it can be avoided. Pain-free will have Y if VAS  $\leq$  1.5 otherwise blank.

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmaceutica | ls (Page ) | X of Y) Protocol: 402-C-414 |
|---|---|---|
| Listing 16.2-8.1: Pc | stsurgical Total Opioid Dose (OMED | mg) and Ofree Status - All Randomized Subjects |
| | 0 to ≤72 hrs or at | hospital |
| Subject | discharge | Opioid-Free |
| XXX-YYYY | XXXX.X | NO |
| XXX-YYYY | _ | YES |

Total dose is dose from end of surgery through timepoint.

Note to programmer: If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y)
Listing 16.2-8.2: Postsurgical Opioid Dosing - All Randomized Subjects

| TREATMEN | T: treatment-name | | | | · | | · | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Time | | | | | Frequency | | Reason | for |
| | | to | | | | Dose | | | Use | |
| | | Dosing | | Dose | Conversion | (OMED | | | | |
| Subject | Date and Time | (hr) | Medication | (units) | Factor | mg) | | Route | | |
| XXX- | | | | | | | XXX | | XXXXXXX | |
| YYYY | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | (XXXXX) | X.XX | XXX.X | | XXXXXXX | | |
| | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | (XXXXX) | X.XX | XXX.X | Xxx | XXXXXXX | XXXXXXX | |
| | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | (XXXXX) | X.XX | XXX.X | Xxx | XXXXXXX | XXXXXXX | |
| | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXXX | (XXXXX) | X.XX | XXX.X | Xxx | XXXXXXX | XXXXXXX | |

Time to Postsurgical Opioid Dosing is time from end of surgery to Postsurgical Opioid medication dose.

**Note to programmer:** If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y)

Listing 16.2-9: Prescription Daily Pain Medication - All Randomized Subjects

TREATMENT: treatment-name

| Subject | Date and Time | Time to<br>Dosing (hr) | Medication | Dose<br>(units) | Route |
|---|---|---|---|---|---|
| XXX-YYYY | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXX | (XXXXX) | XXXXXXX |
| | DDMONYYYYTHH:MM | XXX.X | XXXXXXXXXX | (XXXXX) | XXXXXXX |
| | DDMONYYYYTHH:MM<br>DDMONYYYYTHH:MM | XXX.X<br>XXX.X | XXXXXXXXXXXX | (XXXXX)<br>(XXXXX) | XXXXXXX<br>XXXXXXX |

Time to dosing is time from end of surgery to pain medication dose.

Note to programmer: If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-10: Rescue Mediation - All Randomized Subjects

TREATMENT: treatment-name

| Subject | Date and Time | Time to<br>Dosing (hr) | Medication | Dose<br>(units) | Route |
|---|---|---|---|---|---|
| XXX-YYYY | DDMONYYYYTHH: MM | XXX.X | XXXXXXXXXXX<br>XXXXXXXXXXX | (XXXXX) | XXXXXXX |
| | DDMONYYYYTHH:MM<br>DDMONYYYYTHH:MM<br>DDMONYYYYTHH:MM | XXX.X<br>XXX.X<br>XXX.X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (XXXXX)<br>(XXXXX)<br>(XXXXX) | XXXXXXX<br>XXXXXXX<br>XXXXXXX |

Time to rescue dosing is time from end of surgery to rescue medication dose.

Note to programmer: If medication is 'Other', text should read 'Other: specify-text'. Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-11: Opioid Related Symptom Distress Scale (ORSDS) - All Randomized Subjects

| | nt: trea | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subjec<br>t | Date<br>(Day) | and | Time | Time point | Question | Symptoms | Answer | Score |
| XXX-<br>YYYY | DDMONY<br>(XX) | ҮҮҮТНН | : MM | 24 hrs | Fatigue | Frequency<br>Severity | Rarely<br>Slight | 1<br>1 |
| | | | | | | Bothersomeness | Not at all<br>Average | 1<br>1 |
| | | | | | Drowsiness | Frequency<br>Severity<br>Bothersomeness | Occasionally<br>Severe<br>Very Much | 2<br>3<br>5 |
| | | | | | Inability t<br>Concentrate Nausea | o<br>Frequency<br>Severity<br>Bothersomeness | Average | 3.3 |
| | | | | | | | Composite Score | |

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmaceuti<br>Listing 16.2-12.1: | cals (Page X of Y) Recovery from Caesarean Section Scale (RCSS) - Question Text | Protocol: 402-C-414 |
|---|---|---|
| Question No. | Question Text | |
| 1 | I recovered quickly from my caesarean | |
| 2 | I was able to get out of bed soon after my caesarean | |
| 3 | My mobility was seriously affected by the caesarean | |
| 4 | The caesarean interfered with my ability to care for my baby | |
| 5 | The caesarean prevented me from feeding my baby | |
| 6 | I was able to change my baby soon after the caesarean | |
| 7 | I was able to care for my own hygiene needs soon after surgery | |
| 8 | The pain from the surgery prevented me from doing what I wanted | |
| 9 | I was red for a long home after surgery | |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Listing 16.2-12.2: Recovery from Caesarean Section Scale (RCSS) - All Randomized Subjects

| TREATMENT: | : treatment-name | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Assessment | | | | Question | | | | | | | | | |
| | | | Actual | Deviation | | | | | | | | | | Total |
| Subject | Date and Time (Day) | Scheduled | (hrs) | (hrs) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | Score |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | 72 hrs | XX.X | XX.X | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | XX |
| | DDMONYYYYTHH:MM (XX) | Early Discharge | XX.X | XX.X | Х | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | XX |

Note to programmer: Sort by date and time within subject.

### 402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Protocol: 402-C-414

Listing 16.2-13: Modified Post-Anesthesia Discharge Scoring System (MPADSS) - All Randomized Subjects

TREATMENT: treatment-name

| | Assessment | Qu | Question | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Date and Time (Day) | Schedule<br>(hrs) | Actual<br>(hrs) | Deviation<br>(hrs) | 1 | 2 | 3 | 4 | 5 | Total<br>Score |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | 24 | XX.X | XX.X | X | Х | Х | Х | Х | XX |
| | DDMONYYYYTHH:MM (XX) | 48 | XX.X | XX.X | X | Χ | Χ | Χ | Χ | XX |

Total score = sum of scores.

#### Question:

- 1. Vital signs:  $2 = \le 20\%$ ; 1 = 20-40%; 0 = >40% of preoperative value.
- 2. Ambulation: 2 = steady gait/no dizziness; 1 = with assistance; 0 = none/dizziness
- 3. Nausea and Vomiting: 2 = minimal; 1 = moderate; 0 = severe
- 4. Pain: 2 = minimal; 1 = moderate; 0 = severe
- 5. Surgical bleeding: 2 = minimal; 1 = moderate; 0 = severe

**Note to programmer:** Sort by date and time within subject.

## 402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-14.1: Surgical Fear Questionnaire (SFQ) - Question Text

| Question No. | Question Text |
|---|---|
| 1 | I am afraid of the operation |
| 2 | I am afraid of the anesthesia |
| 3 | I am afraid of the pain after the operation |
| 4 | I am afraid of the unpleasant side effects (like nausea) after the operation |
| 5 | I am afraid my health will deteriorate because of the operation |
| 6 | I am afraid the operation will fail |
| 7 | I am afraid that I won't recover completely from the operation |
| 8 | I am afraid of the long duration of the rehabilitation after the operaon |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-14.2: Surgical Fear Questionnaire (SFQ) - All Randomized Subjects

| TREATMENT: | treatment | -name | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Assessment | | | | | | est | ior | 1 | | | | | |
| | Date an | d Time | | Actual | Deviation | | | | | | | | | Total |
| Subject | (Day) | | Scheduled | (hrs) | (hrs) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Score |
| XXX-YYYY | DDMONYYYY<br>(XX)<br>DDMONYYYY<br>(XX) | | 72 hrs<br>Early<br>Discharge | xx.x<br>xx.x | xx.x<br>xx.x | | X | | | | | | | XX<br>XX |

Note to programmer: Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-15: Pulse Oximetry (Log Form) - All Randomized Subjects

TREATMENT: treatment-name

| Subject | Date and Time | Time Point | Oxygen Saturation (%) |
|----------|-----------------|------------|-----------------------|
| | | | XX.X |
| XXX-YYYY | DDMONYYYYTHH:MM | 0 hr | |
| | | 1 hr | XX.X |
| | | 2 hrs | XX.X |
| | | 3 hrs | XX.X |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Listing 16.2-16: Subject Satisfaction with Post-Surgical Pain Control at 72 hours - All Randomized Subjects

Treatment: treatment-name

| Subject | Date and Time (Day) | Rating | Score |
|---|---|---|---|
| XXX-YYYY | DDMONYAYAMIII MM (VXX) | DVEDENDI V. DI COMPICEI D | 1 |
| | DDMONYYYYTHH:MM (XX) | EXTREMELY DISSATISFIED | 1 |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | DISSATISFIED | 2 |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | NEITHER SATISFIED NOR DISSATISFIED | 3 |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | SATISFIED | 4 |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | EXTREMELY SATISIFIED | 5 |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | EXTREMELY SATISIFIED | 5 |

Note to programmer: Sort by date and time within subject.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-17: Day 14 Phone Call - All Randomized Subjects

TREATMENT: treatment-name

| | | | | No. | of Pain- | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Relate | d | | | | |
| | Day 14 Phor | ne Call | | Unsche | duled | | | | |
| | | | | | | | No. of Hosp<br>Readmission | | Currently Taking<br>Opioid Pain |
| | Schedule A | Actual | Deviation | Phone | | No. of ER | | AE | |
| Subject Date | (days) | (days) | (days) | Calls | Visits | Visit | | Assessed | |
| | | | | | | | | | Y |
| XXX-YYYY DDMONY | YY 1 <b>4</b> | XX.X | XX.X | XX | XX | XXXX | XXXX | Y | |
| | | | | | | | | | N |
| XXX-YYYY DDMONY | YY 1 <b>4</b> | XX.X | XX.X | XX | XX | XXXX | XXXX | Y | |
| | | | | | | | | N | Y |
| XXX-YYYY DDMONY | YY 1 <b>4</b> | XX.X | XX.X | XX | XX | XXXX | XXXX | | |

Note to programmer: If the leading question "were there any ..." is No, then "No. of ..." is 0.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-18: Vital Signs Assessment - All Randomized Subjects

TREATMENT: treatment-name

| | | | | | Heart R | ate | Blood P | ressure ( | mmHg) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Assessment | | | | (bpm) | | Systolic | | Diastol | ic |
| Subject | Date and Time | Schedule<br>(hrs) | Actual<br>(hrs) | Dev.<br>(hrs) | Actual | Change | Actual | Change | Actual | Change |
| XXX-YYYY | DDMONYYYYTHH:MM | Screening | - | - | XX | - | XXX | - | XX | _ |
| | DDMONYYYYTHH:MM | OR | - | - | XX | XX | XXX | -X | XX | X |
| | DDMONYYYYTHH:MM | PACU | XXX.XX | XXX | XX | -XX | XXX | X | XX | -X |
| | DDMONYYYYTHH:MM | 12 hr | XXX.XX | XXX | XX | -XX | XXX | X | XX | -X |
| | DDMONYYYYTHH:MM | 24 hr | XXX.XX | XXX | XX | -XX | XXX | X | XX | -X |
| | DDMONYYYYTHH:MM | 48 hr | XXX.XX | XXX | XX | -XX | XXX | Χ | XX | -X |
| | DDMONYYYYTHH:MM | 72 hr | XXX.XX | XXX | XX | -XX | XXX | X | XX | -X |

<sup>\*=</sup>out of window

Change is change from baseline (Preop).

@=potentially clinically significant value

Protocol: 402-C-414

**Note to programmer:** Sort by Date and time within subject. An asterisk (\*) will be placed next to the deviation if an assessment is out of window. See Table of Time and Events for windows.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-19: Electrocardiogram Findings at Screening - Investigator Assessment - All Randomized

Subjects

Treatment: treatment-name

| Subject | Date and Time | Date | Time | Finding |
|---|---|---|---|---|
| XXX-YYYY | DDMONYYYYTHH:MM | | | Normal |
| XXX-YYYY | DDMONYYYYTHH:MM | | | Abnormal, clinically significant |
| XXX-YYYY | DDMONYYYYTHH:MM | | | Abnormal, not clinically significant |
| XXX-YYYY | DDMONYYYYTHH:MM | | | Normal |
| XXX-YYYY | DDMONYYYYTHH:MM | | | Normal |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Listing 16.2-20: Pain Intensity Scale - Timepoint Questions - All Randomized Subjects

Treatment: treatment-name

Timepoint at Which Subjects was Asleep

| Subject | 12 hrs | 24 hrs | 48 hrs | 72 hrs |
|----------|--------|--------|------------|---------|
| XXX-YYYY | Yes | Yes | Yes | Yes |
| | No | No | No | No |
| | | Yes | Unknown | Unknown |
| | | 100 | Olikilowii | OHAHOWH |

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y)
Listing 16.2-21: Assessment of Itching - All Randomized Subjects

Treatment: treatment-name Itching Any Severity at Screening Visit Visit? Date/Time Subject Itching\* Reason Not Done 0 XXX-YYYY Screening DDMONYYYYTHH:MM XXXXXXXXXXXXXXXXXXXXXX Day 1 No DDMONYYYYTHH:MM 1 XXXXXXXXXXXXXXXXXXXXXX Day 1-3 Yes 2 DDMONYYYYTHH:MM XXXXXXXXXXXXXXXXXXXXXX 3 No DDMONYYYYTHH:MM XXXXXXXXXXXXXXXXXXXXXX Yes DDMONYYYYTHH:MM 10 XXXXXXXXXXXXXXXXXXXX

<sup>\*= 0=</sup> No Itching and 10= Worst Itch

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y) Listing 16.2-22.1: All Adverse Events - All Randomized Subjects

Treatment: treatment-name

| Subject | TEAE | Data Type | Data |
|----------|------|-----------------------------|---------------------------|
| XXX-YYYY | N | Start (Day) | DDMONYYYYTHH:MM (XX) |
| | | Stop (Day) | DDMONYYYYTHH:MM (XX) |
| | | AE Number | X |
| | | System Organ Class | XXXXXXXXXXXXXXX |
| | | Preferred | XXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXXXX |
| | | Severity | XXXXXXX |
| | | Relationship to Study Drug | XXXXXXX |
| | | Action Taken | XXXXXXXXXXXXXXXXX |
| | | Outcome | XXXXXXXXXXXX |
| | | Serious<br>Serious Cause(s) | Yes/No<br>Hospitalization |
| | | AE of Special Interest | Yes/No |

TEAE: Treatment-emergent AE (Y=TEAE/N=Not TEAE)

**Note to programmer:** If AE is ongoing, put ONGOING in stop row. Do not split an AE across pages. Insert a page break between subjects. Use this mock-up for the following listings:

Listing 16.2-22.2: Treatment-emergent Adverse Events - All Randomized Subjects

Listing 16.2-22.3: All Serious Adverse Events - All Randomized Subjects

Listing 16.2-22.4: Treatment-emergent Adverse Events of Special Interest - All Randomized Subjects

402-C-414 (C-section TAP) Statistical Analysis Plan

XXXXXXXXXXXXXXXXXXX AE # XX (or MH # XX)

Protocol: 402-C-414

Pacira Pharmaceuticals (Page X of Y) Listing 16.2-23.1: Prior Medications - All Randomized Subjects

Frequency

Given for AE or MH?

| Treatment | : treatment- | name | |
|-----------|--------------|-------------------|----------------------|
| Subject | Category | Data Type | Data |
| XXX-YYYY | | Start (Day) | DDMONYYYYTHH:MM (XX) |
| | | Stop (Day) | DDMONYYYYTHH:MM (XX) |
| | | Medication Number | X |
| | | ATC Level 1 | XXXXXXXXXXXXXXX |
| | | ATC Level 2 | XXXXXXXXXXXXXXXXX |
| | | ATC Level 3 | XXXXXXXXXXXXXXXXXXX |
| | | ATC Level 4 | XXXXXXXXXXXXXXXXX |
| | | Preferred Name | XXXXXXXXXXXXXXXXXX |
| | | Verbatim | XXXXXXXXXXXXXXXXX |
| | | Route | XXXXXXX |

XXXXXXXX

ATC=Anatomical therapeutic class

Note to programmer: If medication is ongoing, put ONGOING in stop row. Do not split a medication across pages. Insert a page break between subjects. Values for category column are: CONCOMITANT; SURGICAL/ANESTHESIA; NON-MEDICATION; PRIOR. Use this mock-up for the following listings:

Listing 16.2-23.2: Concomitant Medications - All Randomized Subjects

402-C-414 (C-section TAP) Statistical Analysis Plan

(Page X of Y) Pacira Pharmaceuticals Protocol: 402-C-414

| Treatment | : treatment-name | |
|-----------|--------------------|-----------------------------------------|
| Subject | Data Type | Data |
| XXX-YYYY | Start (Day) | DDMONYYYY (XX) |
| | Stop (Day) | DDMONYYYY (XX) |
| | System Organ Class | XXXXXXXXXXXXXXX |
| | Preferred | XXXXXXXXXXXXXXXXX |
| | History Verbatim | XXXXXXXXXXXXXXXXXXX |
| | Start (Day) | DDMONYYYY (XX) |
| | Stop (Day) | DDMONYYYY (XX) |
| | System Organ Class | XXXXXXXXXXXXXXX |
| | Preferred | XXXXXXXXXXXXXXXXX |
| | History Verbatim | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y)
Listing 16.2-25: Intraoperative Medications - Randomized Subjects

Protocol: 402-C-414

| | | TREATMENT: | treatment-name | | | | |
|---|---|---|---|---|---|---|---|
| Subject | Start Date/Time | End Date/Time | Administered | Name | Dose | Unit | Route |
| XXX-YYYY<br>XXX-YYYY | DDMMYYYY/HH:MM | DDMMYYYY/HH:MM | YES<br>NO | OPIOID-NAME | XXX.XX | (UNITS) | XXXX |

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-26: Study Drug Administration - Randomized Subjects

| | Treatment | | Start | Stop | Total Volume |
|---|---|---|---|---|---|
| Subject | | Date | Time | Time | (mL) |
| XXX-YYYY | Right Study Drug<br>Left Study Drug | DDMONYYYY | нн:ММ | нн:мм | XXX |

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-27: Standard of Care - Randomized Subjects

| Subject | TAP Performed/Medication | Date | Start<br>Time | Dose (Unit) |
|---|---|---|---|---|
| XXX-YYYY | Yes/XXXXXX<br>No | DDMONYYYY | нн:мм | Xxxxxx (xxx) |

402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-28: Physical Examination - Randomized Subjects

TREATMENT: treatment-name

| Subject | Date/Time | Body System | Findings | Details<br>Abnormal | if<br>Reason Not Done |
|---|---|---|---|---|---|
| XXX-YYYY | DDMONYYYY | HH:MM | XXX | XXX | XXX |

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414

Listing 16.2-29: Urine Drug Screen, Alcohol Blood Test and Pregnancy Test - All Subjects

| eatment-name | | | | |
|---|---|---|---|---|
| | | Blood | | |
| Visit | Urine Drug | Alcohol | Pregnancy | |
| Screening | XXXXXXX | XXXXXXX | XXXXXXX | |
| Screening | XXXXXXX | XXXXXXXX | XXXXXXX | |
| Screening | XXXXXXX | XXXXXXXX | XXXXXXX | |
| Screening | XXXXXXX | XXXXXXXX | XXXXXXX | |
| | Visit Screening Screening Screening | Visit Urine Drug Screening XXXXXXXX Screening XXXXXXXX Screening XXXXXXXX | Visit Urine Drug Blood Alcohol Screening XXXXXXXXX XXXXXXXX Screening XXXXXXXXX XXXXXXXX Screening XXXXXXXXX XXXXXXXX | Visit Urine Drug Blood Alcohol Pregnancy Screening XXXXXXXXX XXXXXXXXX Screening XXXXXXXXX XXXXXXXXX Screening XXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXX |

### 402-C-414 (C-section TAP) Statistical Analysis Plan

Protocol: 402-C-414

Pacira Pharmaceuticals

(Page X of Y)

Listing 16.2-30: Admission and Discharge - Randomized Subjects

TREATMENT: treatment-name

| | Date and Time (Day) | | |
|---|---|---|---|
| Subject | Admission to Surgical Facility | Admission to PACU | Discharge to PACU |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) |
| XXX-YYYY | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) | DDMONYYYYTHH:MM (XX) |

Total score = sum of scores.

- 1) Vital signs:  $2 = \le 20\%$ ; 1 = 20-40%; 0 = >40% of preoperative value.
- 2) Ambulation: 2 = steady gait/no dizziness; 1 = with assistance; 0 = none/dizziness
- 3) Nausea and Vomiting: 2 = minimal; 1 = moderate; 0 = severe
- 4) Pain: 2 = minimal; 1 = moderate; 0 = severe
- 5) Surgical bleeding: 2 = minimal; 1 = moderate; 0 = severe

402-C-414 (C-section TAP) Statistical Analysis Plan

Listing 16.2-31: Important Protocol Deviations - Randomized Subjects

| TREAT | TREATMENT: treatment-name | | | | |
|---|---|---|---|---|---|
| Site | Subject | Date (day) | Epoch | Deviation Code | Description |
| XXX | XXX-YYYY | DDMONYYYY (XX) | XXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Note to programmer: Subjects may have multiple deviations. Sort deviations by subject and date.

Select DVDECOD, eg, "Restricted Medications Taken", "Non-Compliance/Ultrasound", "Primary Efficacy Assessments", "Other Important Deviations", "Improper Informed Consent Procedure" as specified by the sponsor.

402-C-414 (C-section TAP) Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-414 Listing 16.2-32: Ultrasound Collection - Randomized Subjects

TREATMENT: treatment-name

| | | Ultrasound Image/Vide | eo captured of the TAP<br>ydrodissection | Ultrasound Image/Video captured of<br>the TAP needle placement after study<br>drug infiltration | |
|---|---|---|---|---|---|
| Subject | Ultrasound Guidance used<br>to perform TAP needle<br>placement/Reason if No | regire brac, reason in | Left Side/ Reason if No | Right Side/ Reason if No | Left Side/ Reason if No |
| XXX-YYYY<br>XXX-YYYY | Yes<br>No/xxxxxxx | Yes<br>No/xxxxxx | Yes<br>No/xxxxxx | Yes<br>No/xxxxxx | Yes<br>No/xxxxxx |

402-C-414 (C-section TAP) Statistical Analysis Plan

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-327 |
|---|---|---|
| Listing 16.2-33: Unique Adverse | Events Terms and Associated Coded Terms | |
| MedDRA Terms | | |
| SOC | | |
| Preferred Term | Verbatim(s) | |
| SOC1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| PT1.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXX | |
| PT1.2 | xxxxxxxxxxxxxxxxxxxxxxxx | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX | |
| SOC2 | | |
| PT2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |

Coded using MedDRA v21.1.

Note to programmer: Sort by SOC and preferred term in alphabetical order

402-C-414 (C-section TAP) Statistical Analysis Plan

| | · | |
|---|---|---|
| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-32 |
| Listing 16.2-34: Unique Medication | Terms and Associated Coded Terms | |
| Who Drug Dictionary Terms | | |
| ACT1 | | |
| ACT2 | | |
| ACT3 | | |
| ACT4 | | |
| Preferred name | Verbatim(s) | |
| ATC1 | | |
| ATC1.2 | | |
| PN1.2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX | |
| PN1.2.2 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| ATC2 | | |
| ATC2.2 | | |
| ATC2.3 | | |
| ATC2.4 | | |
| PN2.2.3.4.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |

Coded using WHO Drug Dictionary September 2018.

Note to programmer: Sort by ATC1, ATC2, ATC3, ATC4 and preferred name in alphabetical order

402-C-414 (C-section TAP) Statistical Analysis Plan

# **18 LIST OF FIGURES**

FIGURE 1: MEAN (+/- 95% CI) OF VAS GENERAL PAIN INTENSITY OVER TIME - EFFICACY 139 ANALYSIS SET

FIGURE 2: MEAN (+/- 95% CI) OF VAS INCISION SITE PAIN INTENSITY OVER TIME - EFFICACY ANALYSIS SET 139

402-C-414 (C-section TAP) Statistical Analysis Plan

Figure 1: Mean (+/- 95% CI) of VAS General Pain Intensity Over Time - Efficacy Analysis Set

Figure 2: Mean (+/- 95% CI) of VAS Incision Site Pain Intensity Over Time - Efficacy Analysis Set

Programming note: include all scheduled VAS pain scores